| C | |
|----|---|
| Ц | ٦ |
| C | 5 |
| Č | 2 |
| Č | 5 |
| | ī |
| Ц | ٦ |
| т | _ |
| | _ |
| C | - |
| Ċ | Ľ |
| ĺ | ٠ |
| _ | |
| | _ |
| C | _ |
| ۲ | ١ |
| C | |
| c | _ |
| ŭ | ξ |
| č | 4 |
| | ī |
| ^ | |
| 'n | ^ |
| ÷ | _ |
| | ı |
| ç | 1 |
| C | |
| ú | ٢ |
| Ĺ | ĺ |
| ۵ | |
| | ı |
| C | ) |
| ū | |
| C | - |
| | ı |
| ٢ | • |
| 0 | ٢ |
| T | |
| _ | ١ |
| 2 | Ľ |
| C | 2 |
| Ц | Ĺ |

| Sponsor: | BIOTRONIK SE & Co KG |
|---|---|
| Study name / EAC code: | BIO Guard-MI / HS058 |
| Version and date of the Statistical Analysis Plan: | Version 3.0 from 03Feb2022 |
| Version and date of the underlying Clinical Investigation Plan: | Version 7.0 from 06Apr2021 |

| Print Name & Title | Signature | Date of Signature<br>(DD MMM YYYY) |
|---|---|---|
| Project Manager<br>Sascha Mrosk<br>BIOTRONIK SE & Co. KG<br>Center for Clinical Research<br>Woermannkehre 1<br>D-12359 Berlin | esigned by S. Mrosk<br>on 03. Feb 2022 | 03. Feb 2022 |
| Senior Clinical Scientist Dr. Jürgen Schrader BIOTRONIK SE & Co. KG Center for Clinical Research Woermannkehre 1 D-12359 Berlin | e-signed J Schrader 03 Feb 202 | 03 Feb 2022<br>22 |
| Biostatistician Dr. Bernd Brüsehaber BIOTRONIK SE & Co. KG Center for Clinical Research Woermannkehre 1 D-12359 Berlin | e-signed by Bernd Brüsehaber<br>on 03 Feb 2022 | 03 Feb 2022 |

In this document, the following content is blackend:

1) Pseudo-code



# **Table of Content**

| | ange nistory | 5 |
|---|---|---|
| | on 1.0 | 5 |
| Versi | on 2.0 | 5 |
| Versi | on 3.0 | 6 |
| 1. Int | roduction | 7 |
| 1.1. | Aim | 7 |
| 1.2. | General information | 7 |
| 1.3. | Data for which quality control is required | 8 |
| | Unblinding | |
| 2. Ob | jectives | 9 |
| | vestigational Device | 9 |
| 4. De | | 10 |
| | neral Statistical Procedures | 13 |
| | Descriptive analyses | |
| | nal – dichotomous data (example with dummy data) | 13 |
| | nal data – more than two categories (example with dummy data) | 13 |
| | / metric data (example with dummy data) | 14 |
| | al data | 14 |
| | Significance level | |
| 5.3. | Missing Data | 16 |
| 5.5. | Exclusion of data from confirmatory data analysis | 16 |
| | terim analyses of the primary endpoint (NOTE: Not relevant for the final analyses | |
| 5.6. | Subgroups | |
| | roups CHADS2 | 10<br>19 |
| | roups other | 20 |
| 5.7. | Phase1: Event rate check (NOTE: Not relevant for the final analysis) | |
| 5.8. | Phase2: Interim analyses (NOTE: Not relevant for the final analysis) | |
| 5.9. | Phase2: Final analysis | |
| 5.10. | Analysis software | |
| | ndomization & specific Study Dates | 23 |
| 6.1. | Randomization | |
| 6.2. | Enrollment date | |
| 6.3. | | |
| 6.4. | Initial and latest implantation date | |
| _ | Effective randomization date for the ITT analyses | |
| 6.5. | Effective randomization date for the PP analyses | |
| 6.6. | Final date for the interim ITT analyses (NOTE: Not relevant for the final anal | yisis) |
| 1 0+ 10 | 25 | 25 |
| | Iterim analysis | 25 |
| | Final date for the final PP analyses | |
| 6.8. | Termination Date (= censoring date for the final ITT analyses) | |
| | alysis Sets | 29 |
| | ITT Analysis Set | |
| 7.2. | | |
| | ta for a CONSORT diagram and "study realization" | 32 |
| 8.1. | Enrollment | |
| 8.2. | Termination | _ |
| | seline Data | 33 |
| | Analysis set | |
| | Variables | |
| | Iment | 33 |
| Basel | | 33 |
| | arameter | 35 |
| Medic | | 35 |
| 9.3. | Treatment of Missing and Spurious Data | 36 |

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



| 9.4.<br>9.5. | Exclusion of Particular Information | |
|---|---|---|
| 9.5.<br>9.6. | Hypotheses & Statistical Tests | |
| | <b>,</b> 1 | .30<br>37 |
| | | 45 |
| 11.1. | Analysis set | |
| 11.1. | Variables | |
| | bles for the ITT analysis set | .43<br>46 |
| | bles for the fire analysis set bles for the per-protocol analysis set | 46 |
| 11.3. | Treatment of Missing and Spurious Data | _ |
| 11.4. | Exclusion of Particular Information | |
| 11.5. | Descriptive Analyses | |
| 11.6. | Hypotheses & Statistical Tests | .47<br>17 |
| | | 48 |
| 12.1. | Analysis set | _ |
| 12.1. | Variables | |
| 12.2. | Treatment of Missing and Spurious Data | |
| 12.3. | Exclusion of Particular Information | |
| 12.4. | Descriptive Analyses | |
| 12.5.<br>12.6. | | |
| | Hypotheses & Statistical Testsner sec. EP: Time to all-cause death or heart transpl. | .49<br>50 |
| 13.1. | Analysis set | |
| 13.2. | Variables | |
| 13.3. | Treatment of Missing and Spurious Data | |
| 13.1. | Exclusion of Particular Information | |
| 13.2. | Descriptive Analyses | |
| 13.1. | Hypotheses & Statistical Tests | |
| | · · | 51 |
| 14.1. | Analysis set | |
| 14.2. | Variables | |
| 14.3. | Treatment of Missing and Spurious Data | |
| 14.4. | Exclusion of Particular Information | |
| 14.5. | Descriptive Analyses | |
| 14.6. | Hypotheses & Statistical Tests | |
| | her sec. EP: Time to 1 <sup>st</sup> worsening of the patient status due to heart failure | |
| 15.1. | Analysis set | |
| 15.2. | Variables | |
| 15.3. | Treatment of Missing and Spurious Data | |
| 15.1. | Exclusion of Particular Information | |
| 15.2. | Descriptive Analyses | |
| 15.3. | Hypotheses & Statistical Tests | |
| | , | 54 |
| 16.1. | Analysis set | |
| 16.2. | Variables | |
| 16.3. | Treatment of Missing and Spurious Data | |
| 16.1. | Exclusion of Particular Information | |
| 16.2. | Descriptive Analyses | |
| 16.3. | Hypotheses & Statistical Tests | |
| | , , , | 56 |
| 17.1. | Analysis set | |
| 17.2. | Variables | |
| 17.3. | Treatment of Missing and Spurious Data | |
| 17.1. | Exclusion of Particular Information | |
| 17.2. | Descriptive Analyses | .5/ |
| 17.3. | Hypotheses & Statistical Tests | |
| | | 58 |
| 18.1. | Analysis set | .58 |

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



| 18.2. | Variables | EC |
|---|---|---|
| _ | | |
| 18.3. | Treatment of Missing and Spurious Data | |
| 18.1. | Exclusion of Particular Information | |
| 18.2. | Descriptive Analyses | |
| 18.3. | Hypotheses & Statistical Tests | .59 |
| 19. Otl | ner sec. EP: Time to 1 <sup>st</sup> hosp. resulting from major bleeding | 60 |
| 19.1. | Analysis set | 60 |
| 19.2. | Variables | |
| 19.3. | Treatment of Missing and Spurious Data | |
| 19.1. | Exclusion of Particular Information | |
| _ | | |
| 19.2. | Descriptive Analyses | |
| 19.3. | Hypotheses & Statistical Tests | |
| | | 62 |
| 20.1. | Analysis set | |
| 20.2. | Variables | |
| 20.3. | Treatment of Missing and Spurious Data | 63 |
| 20.1. | Exclusion of Particular Information | 63 |
| 20.2. | Descriptive Analyses | |
| 20.3. | Hypotheses & Statistical Tests | 63 |
| | | 64 |
| 21.1. | Analysis set | _ |
| 21.2. | Variables | |
| 21.2. | | |
| | Treatment of Missing and Spurious Data | |
| 21.1. | Exclusion of Particular Information | |
| 21.2. | Descriptive Analyses | |
| 21.3. | Hypotheses & Statistical Tests | |
| | | 66 |
| 22.1. | Analysis set | |
| 22.2. | Variables | 66 |
| 22.3. | Treatment of Missing and Spurious Data | 67 |
| 22.1. | Exclusion of Particular Information | |
| 22.2. | Descriptive Analyses | |
| 22.3. | Hypotheses & Statistical Tests | |
| | | 68 |
| 23.1. | Analysis set | |
| 23.1. | Variables | |
| 23.3. | Treatment of Missing and Spurious Data | |
| 23.1. | Exclusion of Particular Information | |
| 23.2. | Descriptive Analyses | |
| 23.3. | Hypotheses & Statistical Tests | |
| 24. Otl | | 70 |
| 24.1. | Analysis set | 70 |
| 24.2. | Variables | 70 |
| 24.3. | Treatment of Missing and Spurious Data | |
| 24.1. | Exclusion of Particular Information | |
| 24.2. | Descriptive Analyses | |
| 24.3. | Hypotheses & Statistical Tests | |
| | , · | 72 |
| | Analysis set | |
| 25.1. | | |
| 25.2. | Variables | |
| 25.3. | Treatment of Missing and Spurious Data | |
| 25.1. | Exclusion of Particular Information | |
| 25.2. | Descriptive Analyses | |
| 25.3. | Hypotheses & Statistical Tests | |
| Abbreviat | tions | 74 |



# 0. Change history

#### Version 1.0

Initial document

#### Version 2.0

- General document improvement.
- Aim: Inferential analyses of the endpoints are mandatory to be reported in the final CIR.
- Adaptation to the Clinical Investigation Plan Version (CIP) 6.0.
- Date of discharge from index hospitalization is used as effective randomization date in both groups as defined in the CIP.
- Time to death from any cause or heart transplantation added as secondary endpoint as defined in the CIP
- Chapters for the CONSORT diagram and EQ-5D-5L Questionnaire added.
- History of AF deleted as subgroup because such patients are eligible for the study only in exceptional cases and their number is insufficient for a subgroup analysis.
- Confirmatory analysis of the primary endpoint is tested by a log-rank test stratified by NSTEMI vs. STEMI, which is also used for block randomization.
- Precise definition of the EAEC data, which have been implemented in the CDMS after finalizing SAP version 1-0.
- Precise definition of exclusion of data and censoring date for interim analyses
- Precise definition of primary endpoints based on the data from the EAEC evaluation process considering the open study design.1 This lack of blinding can introduce a bias for several reasons2, which will be prevented by the following procedure: In its initial adjudication, the EAEC classifies the true cause of the event with all available information including BioMonitor data. Next, for any possible endpoint, the most probably adjudication result without BioMonitor information is documented. The analyses of the primary endpoint will be based on this latter adjudication, which is in better accordance with the objective of the study. These changed procedures have been initiated by Steering Committee and Sponsor and approved by the EAEC members and implemented in the EAEC charter.

<sup>-</sup> Example 3: A patient dies in a car accident after he lost control of the vehicle. A post mortem interrogation of the BM shows that the accident occurred after the patient had an episode of ventricular fibrillation. Thus, it is a cardiovascular, not a non-cardiovascular death, as it would be assumed in the control group.



<sup>&</sup>lt;sup>1</sup> The study is conducted in a non-blinded fashion. This is unavoidable due to the fact that the study groups are treated differently with respect to a diagnostic procedure.

In general, more information for the adjudication of endpoints are available in the BioMonitor group. Since the BioMonitor stores information on arrhythmias, it can change the adjudication towards an arrhythmic cause of an event (which would count as primary endpoint), but rarely against it. This asymmetry in available information at the adjudication can change primary endpoints of one type towards another (first example). Then, it would remain without effect on the primary objective of the study, but it would change the distribution of the different kinds of endpoints, with a possible effect on the understanding of the study effect. But as the other two examples show, it can also affect the primary outcome, i.e. it can produce a reduced study effect size:

<sup>-</sup> Example 1: A patient is hospitalized with decompensated heart failure. Only from the BioMonitor it is recognized that atrial fibrillation preceded the heart failure event. In the control group, this would be assumed a heart failure event, but in the BioMonitor group, this would be correctly recognized as an arrhythmia hospitalization.

<sup>-</sup> Example 2 : A patient is hospitalized with general malaise. This is attributed to bradycardia episodes and pauses from the BioMonitor memory (both by the treating investigator and the EAEC). In the control group, this would be probably assumed an "other cardiovascular" event, but in the BioMonitor group, it would be adjudicated as an arrhythmia hospitalization.

#### Version 3.0

- General document improvement, e.g. correction of variable labels and oversights in the previous version
- Information about quality control and unblinding included.
- References to the latest CIP version 7.0, especially the change of the statistical design:
   According to the original statistical planning, the study was designed as a three-stage
   adaptive group sequential test procedure according to O'Brian Fleming with survival
   endpoint, where the inverse normal method is used to combine the separate stage
   information. This strategy is replaced with a single final analysis of all data after study
   termination.Information from the latest version of the CDMS considered for the
   specification of variables derived from raw data.
- Labelling of SAP chapters not relevant for the final analysis.
- Further specification of "major protocol deviations" for the per-protocol analysis.
- More detailed information about the primary endpoint analyses.
- Specification of the variables to be analyzed with respect to the other secondary endpoint "Type of initiated therapies".



# 1. Introduction

#### 1.1. Aim

The aim of this document is to provide detailed instructions for the confirmatory interim analyses of the primary endpoint and on all descriptive and inferential statistical analyses for the final Clinical Investigation Report (CIR). Inferential analyses of the primary and secondary endpoint(s) as defined in this document are mandatory to be reported in the final CIR.

#### 1.2. General information

The text contains verbatim excerpts from the CIP Version 1.0. Such excerpts are italicized with grey background.

The main aspects and the design of the clinical investigation are presented in chapters 2, 3, and 4.

General statistical procedures are summarized in chapter 5. Those methods are used in case there is no other instruction within this document.

Definitions of the specific dates, e.g. effective randomization and termination are presented in chapter 0.

The analysis sets are defined in chapter 7.

Data for the CONSORT diagram and baseline data are handled in chapters 8 and 9.

The primary endpoint is handled in chapters 10 and 11, and the secondary endpoints are handled in the following chapters. Thereby the following statistical considerations are specified:

- Definition of the analysis set for the following analyzes, e.g. excluding patients without any measured or imputed data for this endpoint.
- Definition of the endpoint(s) to be analyzed including references to the source data, e.g.
   CRF sheet and item.
- Treatment of missing and spurious data for evaluation of the above endpoint(s).
- Exclusion of particular information from the evaluation of the above endpoint(s) in addition to the exclusion of patients from the analysis set.
- Statistical alternative hypothesis/hypotheses (HA) to analyze the above endpoint(s).
- Statistical tests intended to analyze the above hypothesis/hypotheses.

In case some variables, which are needed to analyze the pre-specified endpoints, are currently not included in the CDMS, they are indicated with <a href="yellow background">yellow background</a> and the Statistical Analysis Plan (SAP) has to be updated before the first interim analysis or the final analysis.



All variables are defined in tables using the following columns:

| Data file | Name of a data file exported from the CDMS with one data row per unique identifier (e.g. patient-specific "patient_display_ID_full" or event-specific "record_ID"). |
|---|---|
| | A new data file (e.g. "data_SAR") might be generated by merging all relevant data from the original CDMS data files and generating derived variables (e.g. BMI from weight and height or date of first AE episode). |
| Notes | Information whether data has to be presented with descriptive methods as defined in the following sub-chapter, data for listings, or data needed for generating of derived variables only. |
| Variable name | Original name of a variable in the CDMS data file or name of a derived variable (indicated with a suffix "_SAR"). |
| Variable label | Original labels from the CDMS data will be used for generating the SAR unless a new label is defined in this document ("NEW"). |
| | Labels might be omitted or shortened ("") if remaining clear. |
| Variable level | Nominal, ordinal, scale (metric, continuous), or date. |
| Nominal values | Original values from CDMS data will be used for generating the SAR unless new nominal values are defined in this document ("NEW"). |
| | Nominal values might be omitted or shortened ("") if remaining clear. |
| | Nominal values for numeric data this information is not applicable (n.a.). |

# 1.3. Data for which quality control is required

A quality control is needed for analyses of all endpoints(s) as defined in the clinical investigation plan (CIP).

#### 1.4. Unblinding

In the context of the first interim analysis in March 2020, the DSMB discovered inconsistencies in adverse event reporting and consequently recommended unblinding of limited sponsor personnel to perform further investigations on the matter.

For this reason, all persons responsible for SAP 3.0 were unblinded.



# 2. Objectives

#### CIP chapter7.1.1 Primary objectives

The primary objective of the BIO\GUARD-MI study is to investigate whether the early diagnosis of cardiac arrhythmias, provided by the BioMonitor in connection with remote monitoring, and the consequent treatment of the patient will decrease the risk to experience a MACE in patients with a history of MI, CHA2DS2-VASc-Score  $\geq$  4 in men /  $\geq$  5 in women and LVEF > 35 %.

. . .

#### CIP chapter 7.1.2 Secondary objective: Arrhythmia detection

It will be investigated if the implantation of the ICM leads to a faster detection of an arrhythmia that requires a guideline-recommended therapy than a strategy of conventional follow-up.

#### CIP chapter7.1.3 Other secondary objectives

In parallel to the primary objective and the definition of MACE, all individual MACE components will be evaluated separately and compared between the study groups.

- 7.1.3.1 All-cause mortality ...
- 7.1.3.2 Cardiovascular death ...
- 7.1.3.3 Worsening of the patient status due to heart failure ...
- 7.1.3.4 Hospitalization resulting from arrhythmia ...
- 7.1.3.5 Hospitalization resulting from acute coronary syndrome ...
- 7.1.3.6 Hospitalization or death resulting from stroke ...
- 7.1.3.7 Major bleeding requiring hospitalization ...
- 7.1.3.8 Systemic embolism requiring hospitalization ...
- 7.1.3.9 Arrhythmias ...
- 7.1.3.10 Type of initiated therapies ...
- 7.1.3.11 Therapies ...
- 7.1.3.12 Quality of Life (QoL) ...

# 3. Investigational Device

<u>CIP chapter 4.1 Summary description of the investigational device and its intended purpose</u> Investigational device: BioMonitor or CE-approved successor.

The BioMonitor is an ICM used to automatically detect and record episodes of arrhythmia in patients at risk for bradycardia, tachycardia, asystole and AF. The ICM is not intended to deliver any therapy.

The device reports the recorded episodes and the related statistical data via a physician's programmer and telemetrically via BIOTRONIK Home Monitoring.



# 4. Design

#### CIP chapter 8.1 General Considerations

The BIO\GUARD-MI study is a multicenter, prospective, randomized (1:1), controlled, parallel-group, open, international study (including USA) with an event-driven design. The study is operatively divided into 2 phases. In the first phase 640 patients will be enrolled within approximately 2 years after FPI. After 600 patient years of cumulative follow-up have been collected, a blinded analysis will be performed to assess the primary endpoint rate. Based on the assessed rate (see section 11.7), the study will enter the second phase or be discontinued prematurely. This is necessary because it is impossible to obtain solid estimates of the endpoint rates for the included population from the literature. In case of a too low endpoint rate, the study could be expected to fail in its primary objective, even if the BioMonitor group had a much reduced endpoint rate.

In the second phase enrollment will continue in the same way, but in more investigational sites than the first phase, and without interception until up to 2900 patients entered the study. The duration of the second study phase is estimated to last 4 years but ultimately is dependent on when the number of needed endpoints for the final analysis is reached. In the second phase US patients will contribute to the study.

...

## CIP chapter 11.1.1 Group sequential design

According to the original statistical planning, the study was designed as a three-stage adaptive group sequential test procedure according to O'Brian Fleming with survival endpoint, where the inverse normal method is used to combine the separate stage information. This strategy is replaced with a single final analysis of all data after study termination.

The first interim analysis has been performed. The planned second interim analysis will not be done. Due to the O'Brien Fleming design with a very low alpha 1 = 0.00025 for the first interim analysis, an adjusted significance level for the final analysis alpha final = 0.02476 will maintain the global 1-sided significance level alpha = 0.025.



# CIP chapter 8.4.1. CRFs and Forms

Table 2: Overview CRFs and Investigations

| Investigation | ır | a | tion | ge | ne<br>very 6<br>s) | nia<br>form | form | ation | ion |
|---|---|---|---|---|---|---|---|---|---|
| | Enrollment | Baseline | Implantation | Discharge | Telephone<br>contacts (every<br>months) | Arrhythmia<br>notification form | General<br>notification form | IHF notification<br>form | Termination |
| Patient informed consent | Х | | | | | | | | |
| Verification of in- and exclusion criteria | х | | | | | | | | |
| Patient demographics | | X | | | | | | | |
| NYHA class | | X | | | | | | | |
| Echo parameters | | х | | | | | | | |
| Specification of MI | X | | | | | | | | |
| Medical history/Co-<br>morbidities | | x | | | | | | | |
| Cardiovascular medication | | | | X | | | | | |
| Lab parameters | | | | X | | | | | |
| Randomization result | | х | | | | | | | |
| BioMonitor implantation | | | X | | | | | | |
| BioMonitor interrogation | | | X | | | | | | |
| BioMonitor programming | | | x | | | | | | |
| Adverse events | | х | X | X | х | X | Х | х | х |
| Arrhythmia classification | | | | | | Х | | | |
| Evaluation of necessity to contact patient | | | | | | х | х | х | |
| Patient interview | | | | | | X | X | X | |
| Evaluation of necessity of<br>diagnostic procedure | | | | | | x | х | x | |
| Telephone follow-up<br>questionnaire | | | | | x | | | | |
| Quality of life questionnaires | | | | | X | | | | |
| Documentation of: - reason for visit - performed examinations, | | | | | | x | x | x | |
| therapies, modifications | | | | | | | | | |
| Documentation of: - regular or premature termination | | | | | | | | | x |
| - reason for premature<br>termination | | | | | | | | | |

#### CIP chapter 9.1 Overview

Table 3: Study Flowchart

Enrollment

Baseline

Randomization

ICM implantation + Home Monitoring® + "best treatment"

Discharge

Follow up telephone calls every 6 months

Termination



# 5. General Statistical Procedures

## 5.1. Descriptive analyses

#### CIP chapter 11.1.4 Statistical methods

Descriptive analyses: The data are presented using descriptive statistical methods. For metric data sets, the mean values, standard deviation, median, maximum and minimum are stated, if appropriate. Ordinal data are described by the median and interquartile range. For nominal data, absolute numbers and relative frequencies are determined.

For illustration, see the following standard tables with and without subgroup analyses based on dummy data.

#### Nominal - dichotomous data (example with dummy data)

| | | | | Relative |
|--------------------------------|----------|---------|-----------|-----------|
| Variable | | N non- | Absolute | frequency |
| (N total = 10) | Category | missing | frequency | [%] |
| Gender | Female | 9 | 3 | 33.3 |
| History of atrial fibrillation | Yes | 8 | 4 | 50.0 |

| | | | | | Relative |
|---|---|---|---|---|---|
| Variable | | Group | N non- | Absolute | frequency |
| (N total = 10) | Category | Randomization | missing | frequency | [%] |
| Gender | Female | Implant(N group = 4) | 4 | 1 | 25.0 |
| | | Control (N group = 4) | 4 | 2 | 50.0 |
| | | All | 9 | 3 | 33.3 |
| History of atrial fibrillation | Yes | Implant | 4 | 2 | 50.0 |
| | | Control | 4 | 2 | 50.0 |
| | | All | 8 | 4 | 50.0 |

#### Nominal data - more than two categories (example with dummy data)

| Variable | N non- | I | II | II | IV |
|----------------|---------|-----------|-----------|-----------|-----------|
| (N total = 10) | missing | N(%) | N(%) | N(%) | N(%) |
| NYHA class | 8 | 1 (12.5%) | 3 (37.5%) | 3 (37.5%) | 1 (12.5%) |

| Variable | Group | N non- | I | II | II | IV |
|---|---|---|---|---|---|---|
| (N total = 10) | Randomization | missing | N(%) | N(%) | N(%) | N(%) |
| NYHA Class | NYHA Class Implant (N group = 4) | | 0 (0.0%) | 1 (33.3%) | 2 (66.7%) | 0 (0.0%) |
| | Control (N group = $4$ ) | 4 | 1 (25.0%) | 1 (25.0%) | 1 (25.0%) | 1 (25.0%) |
| | All | 8 | 1 (12.5%) | 3 (37.5%) | 3 (37.5%) | 1 (12.5%) |



#### Scale / metric data (example with dummy data)

| Variable | N non- | | | | Lower | | Upper | |
|---|---|---|---|---|---|---|---|---|
| (N total = 10) | missing | Mean | SD | Min | quartile | Median | quartile | Max |
| Age [years] | 9 | 56.1 | 15.9 | 25.0 | 50.0 | 60.0 | 66.0 | 77.0 |
| Weight [kg] | 8 | 78.5 | 13.9 | 55.0 | 69.5 | 78.5 | 89.0 | 99.0 |

| Variable | Group | N non- | | | | Lower | | Upper | |
|---|---|---|---|---|---|---|---|---|---|
| (N total = 10) | Randomization | missing | Mean | SD | Min | quartile | Median | quartile | Max |
| Age [years] | Implant (N group = 4) | 4 | 61.8 | 11.2 | 50.0 | 55.0 | 60.0 | 68.5 | 77.0 |
| | Control (N group = 6) | 4 | 50.3 | 21.5 | 25.0 | 32.5 | 53.0 | 68.0 | 70.0 |
| | All | 9 | 56.1 | 15.9 | 25.0 | 50.0 | 60.0 | 66.0 | 77.0 |
| Weight [kg] | Implant | 3 | 85.0 | 7.0 | 77.0 | 77.0 | 88.0 | 90.0 | 90.0 |
| | Control | 4 | 76.0 | 18.5 | 55.0 | 62.5 | 75.0 | 89.5 | 99.0 |
| | All | 8 | 78.5 | 13.9 | 55.0 | 69.5 | 78.5 | 89.0 | 99.0 |

#### Ordinal data

Identical tables as for metric data but without mean and SD



## 5.2. Inferential analyses

#### CIP chapter 11.1.4 Statistical methods

Inferential analysis of the primary hypothesis: The inverse normal combination test is used to combine the independent increment to a global test statistic. A one-sided logrank test is performed in the context of a confirmatory analysis of the primary hypothesis at every interim and the final analysis.

Explorative multivariable analyses are performed (after the termination of the study, i.e. not after interim analysis) based on the Cox regression model.

Inferential analysis: For the inferential analysis of metric, normal-distributed data, a t-test for interindividual of independent groups or a paired t-test for the intraindividual comparison of paired data is performed. In case the normality assumption of the data is either a priori not justified as specified in the SAP or overtly violated (i.e. by a significant Kolmogorov-Smirnov-Lilliefors or Shapiro-Wilk test result) a non-parametric Wilcoxon-Mann-Whitney rank-sum test or a Wilcoxon-signed-rank test is performed, respectively. For the analysis of relative frequencies, Fisher's exact test is used.

For better comparability of results, a non-parametric Wilcoxon-Mann-Whitney rank-sum test or a Wilcoxon-signed-rank test is performed for all inferential analyses of metric data.

# CIP chapter 11.1.1 Statistical design

According to the original statistical planning, the study was designed as a three-stage adaptive group sequential test procedure according to O'Brian Fleming with survival endpoint, where the inverse normal method is used to combine the separate stage information. This strategy is replaced with a single final analysis of all data after study termination.

The first interim analysis has been performed. The planned second interim analysis will not be done. Due to the O'Brien Fleming design with a very low alpha\_1 = 0.00025 for the first interim analysis, an adjusted significance level for the final analysis alpha\_final = 0.02476 will maintain the global 1-sided significance level alpha = 0.025.

As already specified in SAP 2-0, a stratification for the final analysis of the primary hypothesis is performed for the variable amikind\_multi = STEMI/NSTEMI, which is also used for block randomization.



## 5.3. Significance level

CIP chapter 11.3 Level of significance and the power of the study

The global significance level is of the 1-sided hypothesis is 2.5%.

A statistical power of the final analysis of 80% was used for sample size calculation.

## 5.4. Missing Data

CIP chapter 11.11 Handling of missing, unused and spurious data

Missing data: With respect to the primary hypothesis, drop-outs are considered as censored data and must not be imputed.

Unused data: Data not needed for pre-specified inferential analyzes are minimized and limited to baseline information which can be obtained without any additional burden for the patient. Such data could be used for descriptive and exploratory analyses.

Spurious data are clarified via the query management, i.e. corrected after approval of an investigator. Outliers are identified during the blind review of the data. In case of a clear evidence of a measurement error, the SAP will be updated before breaking the blind in order to avoid any bias.

# 5.5. Exclusion of data from confirmatory data analysis

CIP chapter 11.1.2 Full Analysis set based on the ITT principle

- ... the following patients will be excluded from the analysis set
- Patients of the BioMonitor group and control group in case of a drop-out before discharge from the index hospitalization
- Patients without signed informed consent form

Details are presented in chapter 7.



#### 1st Interim analyses of the primary endpoint (NOTE: Not relevant for the final analysis)

During the course of the study, data may be entered in the CDMS without instantaneous confirmation of the investigator, monitor, or data manager. In any CDMS data export there are record status information for each electronic CRF.

| record_status | record_status_text |
|---------------|----------------------------------------|
| 1 | Completed form |
| 2 | New form |
| 3 | Open issue(s) |
| 1147 | Signed by investigator |
| 1148 | Monitor check in progress, form locked |
| 1149 | Approved by monitor |
| 1150 | Ready for analysis and locked |
| 1151 | Open query |
| 1152 | Answered query |
| 1195 | Adjudication entered |

For the final analysis, all CRFs shall have the status "ready for analysis and locked" or "Adjudication entered" but for the interim analysis some other record\_status values are sufficient as described in the table below. All other CRFs will be excluded from confirmatory data analysis for the interim analysis.

Close before the 1<sup>st</sup> the interim analysis all investigational sites will be intensively monitored to check AE reporting, either to identify AEs which might be classified as primary endpoints or to confirm event-free survival. For obvious reasons, this cannot be done on the same day in all investigational sites. To avoid any bias due to non-monitored data, clinical data occurred after the start date 14JAN2020 of this monitoring phase will be excluded from confirmatory data analysis for the interim analysis.

| CRFs | Sufficient record_status | | Reason |
|---|---|---|---|
| enrollment | | | Monitor check of patient informed consent needed |
| study_termination | , , | , | Monitor check of correct termination date needed |
| discharge<br>adverse_events<br>general_notification<br>arrhythmia_notification<br>who_five_well_being_index<br>eq_5d_5l_questionnaire | 1149, 1150,<br>1152 | window for the interim analysis | Monitor check of clinical data is not needed but event-free survival can be confirmed until the start of the monitoring phase only. |
| baseline | | , | Randomization result is filled in automatically |
| eaec_adjudication <sup>3</sup> | all | all | Quality check via 2-of-3 decisions |

As the investigators have a 14 days period allowed to report Adverse Events, and in reported Adverse Events the querying process and the securing of required documentation for the EAEC takes time, it is not guaranteed that Monitors will not have to return the sites after this "final" day. However, Adverse Events that had an onset after this day will not be used in the analysis.



This document and/or its contents are only for internal use.

## 5.6. Subgroups

#### CIP chapter 11.9 Specification of subgroups

Subgroups are predefined for exploratory analyses with respect to

- the occurrence of the predefined arrhythmias, and to
- the primary endpoint and other predefined outcomes.

All subgroup analyses which are not pre-specified in the chapters 8 or following will be performed as ad-hoc analyses if needed.

# CIP chapter 11.9 Specification of subgroups

The following subgroups are predefined according to their presentation at enrollment:

- All individual components of the CHADS2-score except the age-variable
- Age < median vs. ≥ median
- "Early enrollment" within 40 days of most recent MI vs. "late enrollment" after more than 40 days
- Men vs. women
- CHA2DS2-VASc-score  $\leq 4$  in men  $/ \leq 5$  in women vs.  $\geq 5$  in men  $/ \geq 6$  in women
- LVEF < median vs. ≥ median
- BMI: < 30 vs. BMI ≥ 30</li>
- History of AF yes vs. no
- NSTEMI vs. STEMI
- History or presence of kidney failure yes vs. no

The subgroup "history of AF" defined in the CIP will not be considered for subgroup analyses. This variable is missing in the Baseline CRF because patients with history of atrial fibrillation and a CHADS-VASc score as required by the CIP are indicated to receive oral anticoagulation, which is an exclusion criterion. Thus, patients with history of AF are eligible for the study only in exceptional cases and their number is insufficient for subgroup analyses.



# Subgroups CHADS2

Subgroups with respect to all individual components of the CHADS2 score except the age variable, which is grouped according to the median.

| Data file: Identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_display_id_full | | name | label | level | values |
| data_SAR | descr. | subgroups_chads2_c_SAR4 | Subgroups Congestive Heart Failure | nominal | 0 / 1 |
| data_SAR | descr. | subgroups_chads2_h_SAR <sup>5</sup> | Subgroups hypertension | nominal | 0 / 1 |
| data_SAR | descr. | subgroups_chads2_d_SAR <sup>6</sup> | Subgroups diabetes mellitus | nominal | 0 / 1 |
| data_SAR | descr. | subgroups_chads2_s_SAR <sup>7</sup> | Subgroups stroke or TIA or | nominal | 0 / 1 |
| | | | systematic thromboembolic event | | |







# Subgroups other

Median cut-offs are based on the ITT analysis set.

| Data file: | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| Identifier | | name | label | level | values |
| patient_displ | | | | | |
| ay_id_full | | | | | |
| data_SAR | descr. | subgroups_age_ge_median_SAR <sup>8</sup> | Subgroups age $<$ median (0) vs $\ge$ median (1) | nominal | 0 / 1 |
| data_SAR | descr. | subgroups_mi_enr_ge_41d_SAR9 | Subgroups enrollment after most recent MI $< 41$ days (0) vs $\ge 41$ days (1) | nominal | 0 / 1 |
| data_SAR | descr. | subgroups_gender_SAR <sup>10</sup> | Subgroups gender<br>men (0) vs women (1) | nominal | 0 / 1 |
| data_SAR | descr. | subgroups_cha2ds2vasc_SAR <sup>11</sup> | subgroups CHA2DS2-VASC<br>low (0) vs high (1) | nominal | 0 / 1 |
| data_SAR | descr. | subgroups_Ivef_ge_median_SAR <sup>12</sup> | Subgroups LVEF $<$ median (0) vs $\ge$ median (1) | nominal | 0 / 1 |
| baseline | descr. | subgroups_bmi_ge_30_SAR <sup>13</sup> | Subgroups BMI $<$ median (0) vs $\ge$ median (1) | nominal | 0 / 1 |
| data_SAR | descr. | subgroups_stemi_SAR <sup>14</sup> | Subgroups kind of MI<br>NSTEMI (0) vs STEMI (1) | nominal | 0 / 1 |
| data_SAR | descr. | subgroups_kidney_failure_SAR <sup>15</sup> | Subgroups kidney failure<br>no (0) vs yes (1) | nominal | 0 / 1 |







# 5.7. Phase1: Event rate check (NOTE: Not relevant for the final analysis)

#### CIP chapter 8.1 General considerations

... The study is operatively divided into 2 phases. In the first phase 640 patients will be enrolled within approximately 2 years after FPI. After 600 patient years of cumulative follow-up have been collected, a blinded analysis will be performed to assess the primary endpoint rate. Based on the assessed rate (see section 11.7), the study will enter the second phase or be discontinued prematurely.

..

#### CIP chapter 11.7 Termination Criteria

There is a blinded evaluation of the MACE rates after the event-check, which is no interim analysis because no therapy effect is investigated. If the total number of patients with at least one MACE in both groups is less than 20 patients per 600 patient-years at the end of the event-check phase, the study will be terminated.

. . .

Via the Study News report, Issue 15 from June 2018, the investigators were informed that the gateway to study phase 2 has been reached. The EAEC Board evaluated 20 events as primary endpoint-related. Thus, phase 2 for the study was announced.

## 5.8. Phase2: Interim analyses (NOTE: Not relevant for the final analysis)

#### CIP chapter 8.1 General considerations

In the second phase enrollment will continue in the same way, but in more investigational sites than the first phase, and without interception until up to 2900 patients entered the study.

. . .

The first and second interim analysis will be performed after 124 and 248 primary endpoints, respectively<sup>16</sup>. Within the interim analyses the primary hypothesis will be tested based on the ITT analysis set. Additionally, the stratified randomization procedure will be checked whether there are severe deviations between the BioMonitor and the control group which indicate a failure of the randomization procedure.

No Clinical Investigation Report will be generated. Any person involved in this analysis is obliged to keep all information confidential. The Statistical Analysis Report will be delivered to the DSMB only. The DSMB will inform the steering committee and the sponsor whether to continue the study without any amendments, continue the study with an amendment (e.g. change of the sample size based on the adaptive design), or stop the study for proven superiority according to the O'Brien-Fleming design. The DSMB is also responsible to give recommendations for stopping the study for safety reasons or for futility, if applicable 17.

No other analyses will be conducted for the Statistical Analysis Report which is submitted to the DSMB. Only in case the DSMB recommends the discontinuation of the study, and the Sponsor decides to follow this recommendation, the further procedures will be identical to those specified for the final analysis.



# 5.9. Phase2: Final analysis

CIP chapter 11.2 Sample Size

The original planning assumed that 372 primary events would be required to accept the primary alternative hypothesis with 80% statistical power given an assumed hazard ratio in the population of 0.7452, and the study was to be terminated after this number of endpoints had been collected.

Instead, it was decided to enter the termination phase without any avoidable further delay. Therefore, the intended number of endpoints may not be reached.

After closing the CDMS all analyses specified in this Statistical Analysis Plan have to be performed and a Statistical Analysis Report and a Clinical Investigation Report will be generated.

# 5.10. Analysis software

All analyses are conducted using SAS Version 9.4 for Windows or higher version (SAS Institute Inc., Cary, NC, USA) statistical software.



# 6. Randomization & specific Study Dates

## 6.1. Randomization

| Data file: Identifier | Variable | Variable | Variable | Nominal values |
|---|---|---|---|---|
| patient_display_id_full | name | label | level | |
| Baseline | randassign | Randomization result | nominal | Control (no implant) / Implant |
| data_SAR | rando_SAR <sup>18</sup> | Randomization | nominal | Control / Implant |

#### 6.2. Enrollment date

#### CIP chapter 8.9.5 Point of enrollment and study termination

The point of enrollment is the time at which a patient signs and dates the informed consent form ... Study related procedures, documentation and collection/following of adverse events will start from this day on.

| Data file: Identifier | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| patient_display_id_full | name | label | level | values |
| enrollment | ic date | Date of informed consent (= date of enrollment) | date | n.a. |

# 6.3. Initial and latest implantation date

| Data file:Identifier | Variable | Variable | Variable | Nominal values |
|---|---|---|---|---|
| record_id | name | label | level | |
| implantation | proc_multi | Implantation procedure is | nominal | Initial BioMonitor implantation |
| | | | | BioMonitor exchange |
| implantation | imp_date | Date of implantation | date | n.a. |

| Data file: Identifier | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| patient_display_id_full | name | label | level | values |
| data_SAR | date_initial_implant_SAR19 | Date initial BM implantation | date | n.a. |
| data_SAR | date_latest_implant_SAR <sup>20</sup> | Date of latest BM implantation | date | n.a. |



# 6.4. Effective randomization date for the ITT analyses

CIP chapter 8.2.1 Randomization

. . .

For patients of the BioMonitor group and Control group, the randomization date is defined as the discharge from the index hospitalization.

Time-to-first-event for the ITT analyses start at the effective randomization date<sup>21</sup>.

| Data file: Identifier | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| patient_display_id_full | name | label | level | values |
| discharge | discharge_date | Date of discharge from index hospitalization | date | n.a. |
| data_SAR | date_effrand_ITT_SAR <sup>22</sup> | Date of effective randomization for ITT analysis | date | n.a. |
| | | (discharge from index hospitalization) | | |

# 6.5. Effective randomization date for the PP analyses

CIP chapter 11.1.3 Per-protocol Analysis Set

...

Primary endpoints are not taken into account in the BioMonitor group and in the control group until 1 month after discharge from the index hospitalization.

Time-to-first-event analyzes start at the effective randomization date plus 30 days.

| | - | · | | |
|---|---|---|---|---|
| Data file: Identifier | Variable | Variable | Variable | Nominal |
| patient_display_id_full | name | label | level | values |
| discharge | discharge_date | Date of discharge from index hospitalization | date | n.a. |
| data_SAR | date_effrand_PP_SAR <sup>23</sup> | Date of effective randomization for PP analysis | date | n.a. |
| | | (discharge from index hospitalization) + 30days | | |



 $<sup>^{\</sup>rm 21}$  The term "index hospitalisation" refers to one of the following events:

<sup>-</sup> In patients who are enrolled with an acute myocardial infarction, it is the day on which they are discharged from hospital after conclusion of the treatment for acute myocardial infaction.

<sup>-</sup> In patients who are not enrolled in the context of an acute myocardial infarction, it is they day they leave the physician who enrolled them, with or without implanted device. It is acknowledged that this is not necessarily an overnight hospitalisation but may be a short visit only.

# 6.6. Final date for the interim ITT analyses (NOTE: Not relevant for the final analysis)

# 1st interim analysis

The latest date after index-hospitalization with confirmed information about AEs (see chapter 5.5 is used for censoring for the interim ITT analysis if there is no previous primary endpoint.

| | | , | | |
|---|---|---|---|---|
| Data file: Identifier | Variable | Variable | Variable | Nominal |
| record_id | name | label | level | values |
| general_notification | contact_date | Date of patient contact | date | n.a. |
| general_notification | visit_date | Date of patient visit in investigational site | date | n.a. |
| arrhythmia_notification | contact_date | Date of patient visit in investigational site | date | n.a. |
| arrhythmia_notification | visit_date | Date of patient visit in investigational site | date | n.a. |
| who_five_well_being_index | interview_date | Date questionnaire performed | date | n.a. |
| eq_5d_5l_questionnaire | EQ5D5L_interview_date | Date questionnaire performed | date | n.a. |
| adverse_events | onset_date | Onset date | date | n.a. |
| adverse_events | sae_date | Date AE became serious | date | n.a. |
| adverse_events | end_date | End date of AE | date | n.a. |
| adverse_events | actionhospstart_date | Start date of hospitalization | date | n.a. |
| adverse_events | actionhospend_date | End date of hospitalization | date | n.a. |
| Data file: Identifier | Variable | Variable | Variable | Nominal |
| patient_display_id_full | name | label | level | values |
| discharge | discharge_date | Date of discharge from index hospitalization | date | n.a. |
| study_termination | term_date | Date of study termination | date | n.a. |
| data_SAR | date_final_1interim_SAR <sup>24</sup> | Final date with confirmed information at or after discharge about AEs for the 1st interim analysis (censoring date if there is no | | n.a. |
| | | previous primary endpoint) | | |

# 6.7. Final date for the final PP analyses

#### CIP chapter 11.1.3 Per-protocol Analysis Set

...

Time-to-first-event data are censored after occurrence of

- Cross-overs from the BioMonitor group to the control group or vice versa
- Major protocol violations as defined in section 14.1
- ..

#### CIP chapter 14.1 CIP compliance and exceptions

... A deviation is any failure to follow, intentionally or unintentionally, the requirements of the CIP, including laws, guidelines and other regulation as far as required by the CIP, as well as applicable amendments. Deviations that are likely to seriously affect or that actually have seriously affected the rights or safety or wellbeing of subjects or the scientific integrity of the clinical investigation are major deviations (in the U.S. the term "violation" will be used). Otherwise they are minor deviations (in the U.S. simply referred to as "deviations").

The first major protocol violation will used for censoring for the per-protocol analysis when there is no previous primary endpoint:

- Date of initial implantation<sup>25</sup> in patients randomized to the control group.
- Date of "elective replacement indicator" (ERI) reported on an Arrhythmia Notification CRF, in patients randomized to the BioMonitor group if they do not receive a new device.
- First date of other major protocol violations after the effective randomization date. Major protocol deviations are documented in the CDMS file deviation\_form\_site. None of the events reported here were found to be relevant here except violation of in- an exclusion criteria and cross-overs contrary to randomization. However, these cases will identified by other procedures defined here and this CRF doesn't have to be considered.

<sup>&</sup>lt;sup>25</sup> Note: A patient with implantation before effective randomization PP is not included in the PP analysis set. Thus, the initial implantation date defined here is implicitly defined as implantation after effective randomization PP.



| Data file: Identifier | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| record_id | name | label | level | values |
| eri_form | expl_date | Date of explantation | Date | Yes / No |
| arryhythmia_notification | reason_multi | Reason for assessment | nominal | Arrhythmia/Event notification |
| | | | | ERI notification |
| arryhythmia_notification | helpvar_dateFormCreated | | date | n.a. |

| Data file: Identifier | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| patient_display_id_full | name | label | level | values |
| study_termination | term_date | Date of study termination | date | n.a. |
| data_SAR | date_final_PP_SAR <sup>26</sup> | Date of first major protocol violation after the | date | n.a. |
| | | effective randomization date of the PP analysis or | | |
| | | termination date (censoring date for PP analysis | | |
| | | when there is no previous primary endpoint) | | |





## **6.8. Termination Date (= censoring date for the final ITT analyses)**

CIP chapter 8.9.5 Point of enrollment and study termination

...

Regular point of termination for the individual patient is the respective date of the final study termination visit.

For all non-regular study terminations, the following rules apply:

- In case of patient death, the date of study termination is the date of death.
- In case of HTX, the discharge date from the HTX procedure's hospitalization is the date of study termination.
- In case of withdrawal of consent, the date of study termination is the date of withdrawal of consent.
- If patient is lost to follow-up, the date of termination is the date of last contact of the investigator or of the CRO that collects AEs. Data from the HMSC will not be used to ascertain the vital status of patients for any primary analysis because this might introduce a bias in favor of the BM arm.
- If patient is defined as drop-out patient for any other reason, the date of study termination is the date on which the reason for the drop-out became effective, i.e. the date on which a violation of inclusion criteria was discovered, or on which the investigator excluded the patient for safety reasons.

The variable term\_date compromises the above definition, which is an instruction for the investigator how to report the termination date. The variable term\_date will be checked during monitoring and during the blind review of the data before CDMS freeze or closure.

All remaining patients are terminated when the formal study termination is announced. Therefore, no individual study termination can be later than the formal study termination.

| Data file: Identifier | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| patient_display_id_full | name | label | level | values |
| study_termination | term_date | Date of study termination | date | n.a. |
| study_termination | regular_yn | regular study termination | nominal | Yes / No |



# 7. Analysis Sets

# 7.1. ITT Analysis Set

CIP chapter 11.1.2 Full Analysis set based on the ITT principle

The analysis of the primary hypothesis is performed on the full analysis set based on theintention-to treat (ITT) principle; i.e. the set of data from all randomized patients byminimal and justified elimination of subjects. This set is used to estimate the effect of the experimental intervention with greatest external validity. Subjects allocated to arandomization group are analysed as members of that group irrespective of their compliance to the planned course of treatment, e.g. cross-over to the other group.

The ICH-E9 guideline states that "there are a limited number of circumstances that might lead to excluding randomized subjects from the full analysis set including ... the failure to take at least one dose of trial medication and the lack of any data post randomization."

In accordance to this quideline, the following patients will be excluded from the analysis set

- Patients of the BioMonitor group and control group in case of a drop-out before discharge from the index hospitalization
- Patients without signed informed consent form

| Data file: Identifier | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| patient_display_id_full | name | label | level | values |
| enrollment | ic_yn | Patient has provided written informed consent | nominal | Yes / No |
| study_terminatuion | term_date | Date of study termination | date | n.a. |
| data_SAR | date_effrand_ITT_SAR | Date effective randomization for ITT analysis (discharge from index hospitalization) | date | n.a. |
| data_SAR | analysis_set_itt_SAR <sup>27</sup> | ITT analysis set | nominal | Yes / No |



# 7.2. PP Analysis Set

#### CIP. Chapter 11.1.3 Per-protocol Analysis Set

A supportive analysis of the primary hypothesis is performed on the per-protocol set (efficacy sample), which is a subset of the patients from the above full analysis set who complied sufficiently with the protocol. This set is used to ensure that the data would be likely to exhibit the effects of treatment according to the underlying scientific model.

The Per-Protocol Analysis Set is the subgroup of the Full Analysis set after exclusion of

- Patients with violation of in- or exclusion criteria at enrollment
- Patients with major deviations from the CIP in accordance with the definition given in section 14.1
- Patients of the BioMonitor group without implanted device or drop-out less than 1 month after implantation
- Patients of the control group in case of a drop-out less than 1 month after index hospitalization

#### CIP chapter. 14.1 CIP compliance and exceptions

... A deviation is any failure to follow, intentionally or unintentionally, the requirements of the CIP, including laws, guidelines and other regulation as far as required by the CIP, as well as applicable amendments. Deviations that are likely to seriously affect or that actually have seriously affected the rights or safety or wellbeing of subjects or the scientific integrity of the clinical investigation are major deviations (in the U.S. the term "violation" will be used). Otherwise they are minor deviations (in the U.S. simply referred to as "deviations").

Erroneous, spurious or missing data in a CRF is not a deviation in itself and is handled according to the query processes described in the data management section of this CIP. However, the underlying reason might be a deviation.

Intentional, anticipated deviations from the CIP are only allowed if the deviation is required to protect the subject's rights, safety and well-being or the scientific integrity of the study. In such a case, the investigator will contact the sponsor and obtain prior approval for the deviation. If the deviation occurs in an emergency situation or any other unforeseen situation and is required to protect the patient's life or wellbeing, no prior sponsor approval is required. In case of a study deviation, either anticipated or unanticipated, both the investigator as well as the sponsor may request drop-out/premature study termination of the patient, based on the nature and/or consequences of the deviation.

To be more precise, the per-protocol analysis set<sup>28</sup> is given by the ITT analysis set excluding

- patients with violation of in- or exclusion criteria,
- patients with study termination before the effective randomization date for the PP analyses
- patients randomized to the BioMonitor group without implantation
- patients randomized to the the control group with implantation before the effective randomization date for the PP analyses, and
- patients with other major protocol violations before the effective randomization date.
  Major protocol deviations are documented in the CDMS file deviation\_form\_site. None of
  the events reported here were found to be relevant here except violation of in- an
  exclusion criteria and cross-overs contrary to randomization. However, these cases will
  identified by other procedures defined here and this CRF doesn't have to be considered.

<sup>&</sup>lt;sup>28</sup> Note: Patients with major protocol violations later than 30 days after index discharge are included in the perprotocol analysis set. However, data after the occurrence of the protocol violation is not taken into account (see chapter 6.5).



| Data file: | | 1 | 1 | Nominal |
|---|---|---|---|---|
| | name | label | level | values |
| patient_display_id_full | | | | |
| enrollment | in01_yn, in02_yn, in03_yn, In04_yn | Inclusion criteria | nominal | Yes /No |
| enrollment | ex01_yn, ex02_yn, ex03_yn, | Exclusion criteria | nominal | |
| | ex04_yn, ex05_yn, ex06_yn, | | | |
| | ex07_yn, ex08_yn, ex09_yn, | | | |
| | ex10_yn | | | |
| data_SAR | analysis_set_pp_SAR <sup>29</sup> | Per-protocol analysis set | nominal | Yes / No |



All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



# 8. Data for a CONSORT diagram and "study realization"

This data are analyzed exclusively for the final statistical analysis report. Data are reported for all patients in the complete ITT analysis set as well as separately for the BioMonitor and the control group and for the complete PP analysis set as well as for the BioMonitor and the control group, respectively.

#### 8.1. Enrollment

- Number of patients
- Number of patients per site
- Date of First-Patient-In
- Date of Last-Patient-In

#### 8.2. Termination

- Date of First-Patient-Out
- Date of Last-Patient-Out

•

| Data file:<br>Identifier<br>patient_display<br>_id_full | | Variable<br>name | | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| study_<br>termination | descriptive | , | Regular<br>study<br>termination | nominal | Yes<br>No |
| study_<br>termination | Descriptive<br>for<br>regular_yn<br>= No | multi — | Please<br>indicate the<br>reason<br>for early<br>study<br>termination | | Patient death Withdrawal of patient consent Investigator initiated drop-out Loss to follow-up Early discovery of a violation of inclusion or exclusion criteria Heart transplantation Other |

| Data file: Identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_display_id_ | | name | label | level | values |
| full | | | | | |
| enrollment | Case listings for | ic_date | Date of informed consent | date | n.a. |
| discharge | regular_yn = | discharge_date | Date of discharge from index hospitalization | | |
| study_termination | No | term_date | Date of study termination | | |
| study_termination | | reason_multi | reason for early study termination | nominal | |

| Data file:<br>Identifier<br>patient_display<br>_ id_full | | | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| study_<br>termination | descriptive<br>data<br>including<br>cumulative<br>duration | , – – – – | Days from effective randomization for ITT analysis to termination | metric | n.a. |
| study_<br>termination | descriptive<br>data<br>including<br>cumulative<br>duration | | Days from effective randomization for PP analysis to termination | metric | n.a. |



# 9. Baseline Data

# 9.1. Analysis set

These data are analyzed exclusively for the final statistical analysis report. Data are reported for all patients in the complete ITT analysis set<sup>32</sup> as well as separately for the BioMonitor and the control group and for the complete PP analysis set<sup>33</sup> as well as for the BioMonitor and the control group, respectively.

#### 9.2. Variables

#### **Enrollment**

| Data file: Identifier | Notes | Variable | Variable | | Nominal |
|---|---|---|---|---|---|
| patient_display_id_full | | name | label | level | values |
| baseline | descr. | gender_fm | Gender | nominal | Male / Female |
| baseline | | | | | |
| enrollment | descr. | ami_lma | Left main artery | nominal | True / False |
| enrollment | descr. | ami_lad | Left anterior descending artery (LAD) | nominal | True / False |
| enrollment | descr. | ami_cx | Circumflex artery (CX) | nominal | True / False |
| enrollment | descr. | ami_rca | Right coronary artery (RCA) | nominal | True / False |
| enrollment | descr. | amitreat_pr | Percutaneous revascularization | nominal | True / False |
| enrollment | descr. | amitreat_t | Thrombolysis | nominal | True / False |
| enrollment | descr. | amitreat_0 | NEW: Other kind of MI treatment | nominal | True / False |
| enrollment | descr. | amikind_multi | Kind of MI | nominal | STEMI / NSTEMI |
| enrollment | descr. | amifirst_yn | First occurrence of MI | nominal | Yes / No |
| enrollment | descr. | ami_no | Number of previous MI | metric | n.a. |

#### **Baseline**

| Data file:<br>Identifier<br>patient_display_id<br>_full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| baseline | descr. | | | | |
| baseline | desc. | hidden_age | Age at enrollment | Scale | n.a. |
| baseline | descr. | weight_kg | Weight [kg] | scale | n.a |
| baseline | descr. | height_cm | Height [cm] | scale | n.a. |
| baseline | descr. | bmi | BMI [kg/m2] | scale | n.a. |
| baseline | descr. | bsa | BSA (Mosteller) [m2] | scale | n.a. |
| baseline | no report | lvef_percent | NEW: LVEF after initial AMI treatment [%] | scale | n.a. |
| baseline | no report | lvef_percent_<br>amend1 | NEW: LVEF measurement, performed within 6 months before enrollment [%] | scale | n.a. |
| data_SAR | descr. | lvef_SAR <sup>34</sup> | LVEF (before amendment or -if missing-<br>after amendment) [%] | scale | n.a. |
| baseline | descr. | lav_ml | Left atrial volume [ml] | scale | n.a. |
| baseline | descr. | lvdv_ml | Left ventricular diastolic volume [ml] | scale | n.a. |
| baseline | descr. | lvdvbsa_mlm2 | LVDV/BSA [ml/m2] | scale | n.a. |
| baseline | descr. | lvsv_ml | Left ventricular systolic volume [ml] | scale | n.a. |
| baseline | descr. | lvsvbsa_mlm2 | LVSV/BSA [ml/m2] | scale | n.a. |



| | I | | L | | I |
|---|---|---|---|---|---|
| Data file: Identifier | Notes | | Variable | Variable | Nominal |
| patient_display_id_full | | name | label | level | values |
| baseline | descriptive | Gender_fm | Gender | nominal | Female / Male |
| baseline | | | NEW: Congestive Heart Failure | nominal | Yes / No |
| baseline | | chfnyha_multi | NYHA class | nominal | I / II / III / IV |
| baseline | descriptive | nyha_SAR <sup>35</sup> | NYHA class | ordinal | 1/2/3/4 |
| baseline | descriptive | str_yn | Stroke | nominal | Yes / No |
| baseline | descriptive | tia_yn | Transient ischemic attack | nominal | Yes / No |
| baseline | descriptive | ste_yn | Systemic thromboembolic event | nominal | Yes / No |
| baseline | | | Hypertension | nominal | Yes / No |
| baseline | | | Peripheral artery disease | nominal | Yes / No |
| baseline | descriptive | dia_yn | Diabetes mellitus | nominal | Yes / No |
| baseline | descriptive | vhd_multi | Valvular heart disease | nominal | Yes / No / Not known |
| baseline | with | mca_multi | Myocarditis | nominal | Yes / No / Not known |
| baseline | "Not known " | ren_multi | Renal disease | nominal | Yes / No / Not known |
| baseline | to be | thy_multi | Thyroid dysfunction | nominal | Yes / No / Not known |
| baseline | analyzed | cop_multi | COPD | nominal | Yes / No / Not known |
| baseline | as missing | hep_multi | Hepatic disease | nominal | Yes / No / Not known |
| baseline | data | sle_multi | Sleep apnea | nominal | Yes / No / Not known |
| baseline | descriptive | chads2_SAR <sup>36</sup> | CHADS2 Score | ordinal | 0/1/2/3/4/5/6 |
| data_SAR | descriptive | chads2_SAR <sup>37</sup> | CHADS2 Score (SAR) | ordinal | 0/1/2/3/4/5/6 |
| baseline | descriptive | cha2ds2vasc <sup>38</sup> | CHA2DS2-VASc-Score | ordinal | 0/1/2/3/4/5/6 |
| | | | | | /7/8/9 |
| baseline | descriptive | | CHA2DS2-VASc-Score (SAR) | ordinal | 0/1/2/3/4/5/6 |
| | | SAR <sup>39</sup> | | | /7/8/9 |







# Lab parameter

| Data file: Identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_display_id_full | | name | label | level | values |
| discharge | no report | date_created | Date created | date | n.a. |
| discharge | descriptive | lab1 | Potassium [mmol/I] | scale | n.a. |
| discharge | descriptive | lab2 | Sodium [mmol/I] | scale | n.a. |
| discharge | no report | lab3 | Troponine | scale | n.a. |
| discharge | no report | lab3_multi | Troponine: Specification | nominal | Troponin C (Tn-C) ng/ml |
| | | | | | Troponin I (cTnI) ng/ml |
| | | | | | Troponin T (cTnT) µg/l |
| data_SAR | descriptive | lab3c_SAR <sup>40</sup> | Troponine C [ng/ml] | scale | n.a. |
| data_SAR | | lab3i_SAR <sup>41</sup> | Troponine I [ng/ml] | scale | n.a. |
| data_SAR | descriptive | lab3t_SAR <sup>42</sup> | Troponine T [mue_g/l] | scale | n.a. |
| discharge | descriptive | lab4 | eGFR [ml/min] | scale | n.a. |
| discharge | no report | lab5 | NEW: Haemoglobin | scale | n.a. |
| discharge | no report | lab5_multi | Please specify | | mmol/l |
| | - | | | | g/dl |
| data_SAR | descriptive | lab5_SAR <sup>43</sup> | Haemoglobin [mmol/l] | scale | mmol/l |

# **Medication**

| Data file: Identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_display_id_full | | name | label | level | values |
| discharge | descriptive | concmed01 - | Cardiovascular medication | nominal | Yes/ No |
| | | concmed11 | | | |
| discharge | descriptive | ncconcmed1- | Non-cardiovascular medication | nominal | Yes/ No |
| | | noconcmed4 | | | |
| discharge | case listing for | concmed0911_spec | Please specify (Anticoagulation | text | n.a. |
| | concmed09 = True OR | | treatment Other) | | |
| | concmed11 = True | | | | |

All rights pertaining to this document are exclusively held





## 9.3. Treatment of Missing and Spurious Data

Missing data are not imputed.

Spurious data, which were not clarified by the query process before CDMS closure, are indicated. If appropriate, descriptive and inferential analyses are performed both with /without such data.

#### 9.4. Exclusion of Particular Information

No data from the previous defined analysis set are excluded from the analysis except those defined in chapter 5.5, if applicable.

#### 9.5. Descriptive Analyses

Descriptive data are presented via tables as specified in chapter 5.1.

## 9.6. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses / tests for the baseline data in the CIP.

However, a potential imbalance between BioMonitor and control group with respect to the stratification variable amikind\_multi = STEMI/NSTEMI will be analyzed based on Fisher's exact test. 44

 $<sup>^{44}</sup>$  Even if the randomization procedure will not sufficient and there will be an imbalance amikind\_multi = STEMI / NSTEMI, no bias is expected for the primary endpoint analysis based on the stratified logrank test.


# 10. Pre-processing EAEC data for the primary and secondary endpoints

Each event from the EAEC-adjudication data file is identified by a parent\_record\_id variable. There are at least three data lines per event containing the adjudication of the three board members. In case of deviating decisions of the board members for a specific variable, a 2-of-3 decision is used for further analyses. However, a final adjudication of the chair, which is identified by the variable eac\_complete\_chair = Yes, overrules the evaluations of the other EAEC Members. According to EAEC working procedure, there are at least 2 identical adjudications or a chair decision for each event.

In its initial adjudication, the EAEC classifies the uncorrected<sup>45</sup> cause of the event with all available information including BioMonitor data. Next, for any possible endpoint, the most probably adjudication result without BioMonitor information is documented. The analyses of the endpoints will be based on this variables type\_of\_event\_ae2 and death\_prim\_cause2, which are in better accordance with the objective of the study. However, for the primary endpoint a safety analysis is also performed for the uncorrected variables type\_of\_event\_ae and death\_prim\_cause.

#### CIP Chapter 8.3.1 Primary Endpoint

The primary endpoint is the time from randomization (definition see section 8.2.1) to the first MACE during the clinical investigation. Patients without MACE are censored, i.e. the time from randomization until the earliest date of drop-out, study termination, or date of freezing the Clinical Data Management System database (in case of interim analyses) is considered. Patients who reach the primary endpoint will continue to be followed up until the formal termination of the study is announced (see section 8.1).

A major adverse cardiac event (MACE) comprises the following events:

- Cardiovascular death
- Worsening of the patient status due to heart failure, requiring acute unscheduled hospitalization or urgent visit

or acute unscheduled hospitalization due to adverse events (AE) of the following list:

- Arrhythmia
- Acute coronary syndrome
- Stroke
- Major bleeding
- Systemic embolism

Heart transplantation (HTX) is also a component of "worsening of the patient status due to heart failure, requiring acute unscheduled hospitalization or urgent visit".

<sup>&</sup>lt;sup>45</sup> The "uncorrected" adjudication refers to the assumed true cause of the event after considering of all available information including that coming from the BioMonitor. Because the latter is not available in the control group, this information bias can distort the true treatment effect, and the primary analysis of the treatment effect is based on the adjudication that the EAEC gives und the assumption that no BioMonitor information was available. A detailed justification is given in the EAEC charter.



| Data file:<br>Identifier<br>record_id | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| eaec_<br>adjudication | report | eac_<br>complete_<br>chair | Is chair adjudication for this event applied and complete? | nominal | Yes<br>No |
| eaec_<br>adjudication | No<br>report | type_of_<br>event | Please specify<br>type of event | nominal | Death without prior hospitalisation<br>Heart transplantation<br>Acute unscheduled hospitalisation or urgent HF visit<br>Scheduled hospitalisation or Home Monitoring triggered<br>No hospitalisation / no endpoint due to other reason |
| eaec_<br>adjudication | No<br>report | type_of_<br>event_ae <sup>46</sup> | Primary cause of<br>Unscheduled<br>hospitalisation /<br>urgent visit | nominal | Myocardial infarction Heart failure (urgent visit) Heart failure (hospitalisation) Arrhythmia Stroke Major bleeding Transient ischemic attack Systemic embolism other cardio-vascular non-cardiovascular Undetermined hospitalization or undetermined urgent visit |
| eaec_<br>adjudication | | death_<br>prim_cause | Primary cause of<br>death | nominal | Myocardial infarction Heart failure Sudden cardiac death Stroke Cardiovascular hemorrhage Systemic embolism other cardio-vascular non-cardiovascular undetermined |
| eaec_<br>adjudication | report | date1_<br>of_event | Date of event | date | n.a. |
| eaec_<br>adjudication | report | h | Date of death | date | n.a. |
| eaec_<br>adjudication | | death_<br>occured | Patient death<br>during<br>hospitalization /<br>transplantation | nominal | Yes<br>No |

 $<sup>^{\</sup>rm 46}$  Note new classification "Undetermined hospitalization or undetermined urgent visit"



| Data file:<br>Identifier<br>record_id | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| eaec_<br>adjudication | No<br>report | contribution_<br>significant | The BioMonitor contributed significantly to the adjudication result, so that the result would most probably have been different without the information from the BioMonitor | nominal | Yes<br>No |
| eaec_<br>adjudication | | type_of_<br>event_ae2 | Primary cause of Unscheduled hospitalisation / urgent visit The most probably adjudication result without BioMonitor information would have been | nominal | Myocardial infarction Heart failure (urgent visit) Heart failure (hospitalisation) Arrhythmia Stroke Major bleeding Transient ischemic attack Systemic embolism other cardio-vascular non-cardiovascular |
| eaec_<br>adjudication | | death_<br>prim_cause2 | Primary cause of death The most probably adjudication result without BioMonitor information would have been | nominal | Myocardial infarction Heart failure Sudden cardiac death Stroke Cardiovascular hemorrhage Systemic embolism other cardio-vascular non-cardiovascular undetermined |
| data_eaec_<br>adjudication_<br>SAR | | type_of_<br>event_ae_c <sup>47</sup> | Primary cause of Unscheduled<br>hospitalisation / urgent visit<br>(corrected data) | nominal | Myocardial infarction Heart failure (urgent visit) Heart failure (hospitalisation) Arrhythmia Stroke Major bleeding Transient ischemic attack Systemic embolism other cardio-vascular non-cardiovascular |
| data_eaec_<br>adjudication_<br>SAR | | death_<br>prim_cause_c <sup>48</sup> | Primary cause of death<br>(corrected data) | nominal | Myocardial infarction Heart failure Sudden cardiac death Stroke Cardiovascular hemorrhage Systemic embolism other cardio-vascular non-cardiovascular undetermined |



| Data file: Identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| parent_record_id | | name | label | level | values |
| data_ep_SAR | No | pep_c_2of3chair_SAR <sup>49</sup> | (Corrected) primary EP (based on a 2-of-3 or | nominal | Yes |
| | report | | final chair adjudication of the EAEC) | | No |
| data_ep_SAR | No | pep_u_2of3chair_SAR <sup>50</sup> | Uncorrected primary EP (based on a 2-of-3 or | nominal | Yes |
| | report | | final chair adjudication of the EAEC) | | No |
| data_ep_SAR | No | date_pep_c_2of3chair_SAR <sup>51</sup> | Date of (corrected) primary EP (based on a | date | n.a. |
| | report | | 2-of-3 or final chair adjudication of the EAEC) | | |
| data_ep_SAR | No | | | | n.a. |
| | report | | 2-of-3 or final chair adjudication of the EAEC) | | |

For each triplet eaec\_adjudication variable, an unique composite variable will be generated based on a 2-of-3 or chairman decision. For better readability, the index (\*) is used instead of the index "2of3chair\_SAR", which is used for other derived data.







| Data file: | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| Identifier | | name | label | level | values |
| parent_record_id | | | | | |
| data_ep_SAR | No | death_2of3chair_SAR <sup>53</sup> | All cause death (based on a 2-of-3 or final | nominal | Yes / No |
| | report | | chair adjudication of the EAEC) | | |
| data_ep_SAR | No | | | date | n.a. |
| | report | | chair adjudication of the EAEC) | | |
| data_ep_SAR | No | cvdeath_2of3chair_SAR55 | CV death (based on a 2-of-3 or final chair | nominal | Yes / No |
| | report | | adjudication of the EAEC) | | |
| data_ep_SAR | No | date_cvdeath_2of3chair_SAR56 | Date of HTX (based on a 2-of-3 or final | date | n.a. |
| | report | | chair adjudication of the EAEC) | | |
| data_ep_SAR | No | htx_2of3chair_SAR <sup>57</sup> | HTX (based on a 2-of-3 or final chair | nominal | Yes / No |
| | report | | adjudication of the EAEC) | | |
| data_ep_SAR | No | date_htx_2of3chair_SAR <sup>58</sup> | Date of HTX (based on a 2-of-3 or final | date | n.a. |
| | report | | chair adjudication of the EAEC) | | |







| Data file: | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| Identifier | | name | label | level | values |
| parent_record_id | | | | | |
| data_ep_SAR | No | hf_2of3chair_SAR <sup>59</sup> | Hospitalization or urgent visit for worsening of | nominal | Yes / No |
| | report | | the patient status due to heart failure, or death | | |
| | | | due to heart failure (based on a 2-of-3 or final | | |
| | | | chair adjudication of the EAEC) | | |
| data_ep_SAR | No | date_hf_2of3chair_SAR <sup>60</sup> | Date of hospitalization or urgent visit for | date | n.a. |
| | report | | worsening of the patient status due to heart | | |
| | | | failure, or death due to heart failure (based on a | | |
| | | | 2-of-3 or final chair adjudication of the EAEC) | | |
| data_ep_SAR | No | arr_2of3chair_SAR <sup>61</sup> | hospitalization resulting from an arrhythmia or | nominal | Yes / No |
| | report | | death resulting from arrhythmia (based on a 2- | | |
| | | | of-3 or final chair adjudication of the EAEC) | | |
| data_ep_SAR | No | date_arr_2of3chair_SAR <sup>62</sup> | Date of hospitalization resulting from an | date | n.a. |
| | report | | arrhythmia or death resulting from arrhythmia | | |
| | | | (based on a 2-of-3 or final chair adjudication of | | |
| | | | the EAEC) | | |







| Data file: | | Variable | | Variable | |
|---|---|---|---|---|---|
| Identifier parent_record_id | | name | label | level | values |
| data_ep_SAR | No<br>report | acs_2of3chair_SAR <sup>63</sup> | Hospitalization resulting from acute coronary syndrome or death resulting from acute coronary syndrome. (based on a 2-of-3 or final chair adjudication of the EAEC) | nominal | Yes / No |
| data_ep_SAR | No<br>report | date_acs_2of3chair_SAR <sup>64</sup> | Date of hospitalization resulting from acute coronary syndrome or death resulting from acute coronary syndrome (based on a 2-of-3 or final chair adjudication of the EAEC) | date | n.a. |
| data_ep_SAR | No<br>report | stroke_2of3chair_SAR <sup>65</sup> | Hospitalization resulting from stroke (based on a 2-of-3 or final chair adjudication of the EAEC) | nominal | Yes / No |
| data_ep_SAR | No<br>report | date_stroke_2of3chair_SAR <sup>66</sup> | Date of hospitalization resulting from stroke (based on a 2-of-3 or final chair adjudication of the EAEC) | date | n.a. |







| Data file:<br>Identifier<br>parent_record_id | | Variable<br>name | L 1 1 1 1 1 1 | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| data_ep_SAR | No<br>report | bleed_2of3chair_SAR <sup>67</sup> | hospitalization resulting from major bleeding<br>or death resulting from major bleeding (based<br>on a 2-of-3 or final chair adjudication of the<br>EAEC) | nominal | Yes / No |
| data_ep_SAR | No<br>report | date_bleed_2of3chair_SAR <sup>68</sup> | Date of hospitalization resulting from major bleeding or death resulting from major bleeding (based on a 2-of-3 or final chair adjudication of the EAEC) | date | n.a. |
| data_ep_SAR | No<br>report | emb_2of3chair_SAR <sup>69</sup> | | nominal | Yes / No |
| data_ep_SAR | No<br>report | date_emb_2of3chair_SAR <sup>70</sup> | Date of hospitalization resulting from systemic embolism or death resulting from systemic embolism (based on a 2-of-3 or final chair adjudication of the EAEC) | date | n.a. |





### 11. Primary Endpoint

#### 11.1. Analysis set

Any interim analysis is based on the ITT analysis set.

All analyses for the final statistical analysis report are based on the ITT analysis set<sup>71</sup> and the per-protocol analysis set<sup>72</sup>. Thereby, subgroup analyses are performed for the ITT analysis set only.

#### 11.2. Variables

#### CIP Chapter 8.3.1 Primary Endpoint

The primary endpoint is the time from randomization (definition see section 8.2.1) to the first MACE during the clinical investigation. Patients without MACE are censored, i.e. the time from randomization until the earliest date of drop-out, study termination, or date of freezing the Clinical Data Management System database (in case of interim analyses) is considered. Patients who reach the primary endpoint will continue to be followed up until the formal termination of the study is announced (see section 8.1).

A major adverse cardiac event (MACE) comprises the following events:

- Cardiovascular death
- Worsening of the patient status due to heart failure, requiring acute unscheduled hospitalization or urgent visit

or acute unscheduled hospitalization due to adverse events (AE) of the following list:

- Arrhythmia
- Acute coronary syndrome
- Stroke
- Major bleeding
- Systemic embolism



#### Variables for the ITT analysis set

| Data file: Identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_display_id_full | | name | label | level | values |
| data_SAR | descr. | any_pep_ITT_SAR <sup>73</sup> | Any prim EP occurred at or after | nominal | Yes / No |
| | | | effective randomization ITT | | |
| data_SAR | No | date_1pep_ITT_SAR <sup>74</sup> | Date of 1st prim EP at or after | date | n.a. |
| | report | | effective randomization ITT | | |
| data_SAR | descr. | days_effrand_to_1pep_ITT_SAR <sup>75</sup> | Days from effective randomization | scale | n.a. |
| | | | to first prim EP or censoring ITT | | |

#### Variables for the per-protocol analysis set

| Data file: Identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_display_id_full | | name | label | level | values |
| data_SAR | descr. | | Any prim EP occurred at or after effective randomization PP | nominal | Yes / No |
| data_SAR | No<br>report | | Date of 1st prim EP at or after effective randomization PP | date | n.a. |
| data_SAR | descr. | days_effrand_to_1pep_PP_SAR <sup>78</sup> | Days from effective randomization to first prim EP or censoring PP | scale | n.a. |





Spurious data, which were not clarified by the query process before CDMS closure, are indicated. If appropriate, descriptive and inferential analyses are performed both with /without such data.

#### 11.4. Exclusion of Particular Information

No data from the previous defined analysis set are excluded from the analysis except those defined in chapter 5.5, if applicable.

#### 11.5. Descriptive Analyses

If applicable, mean and median survival times are presented by using the Kaplan-Meier estimates. Kaplan-Meier survival figures are presented for illustration.

Other descriptive data will be presented via tables as specified in chapter 5.1.

#### 11.6. Hypotheses & Statistical Tests

#### CIP Chapter 7.2 Primary hypotheses

For assessing the primary endpoints, Kaplan-Meier curves will be constructed for the time to first MACE for both study groups according to the intention-to-treat principle. The hazard ratio is defined as the rate of the BioMonitor group divided by the rate of the control group.

The following set of hypotheses (null hypothesis H0 and alternative hypothesis HA) will be tested. More detailed information about the endpoints is provided in section 8.3:

- $H_0$ : Null hypothesis:  $H_0$ : HR  $\geq 1$  which means that monitoring patients of the BioMonitor group will not lead to a longer time-to-first-event of MACE compared to the control group.
- $H_A$ : Alternative hypothesis:  $H_A$ : HR < 1 which means that monitoring patients of the BioMonitor group will lead to a longer time-to-first-event of MACE compared to the control group.

It is expected that there is a HR < 1 in favour of the BioMonitor group. A rejection of the null hypothesis indicates that the BioMonitor group has a statistically significant longer time to first MACE event compared to the control group.

The confirmatory analysis of the primary hypothesis is performed according to the methods defined in chapter 0. based on the first primary endpoint after the effective randomization date or censoring at the termination date in the ITT analysis set.

The test of the primary hypothesis is repeated according to the methods defined in chapter 0. based on the first endpoint after the effective randomization date for the PP analysis or censoring at the final date for the final PP analyses in the PP analysis set.

In case the primary alternative hypothesis can be accepted, hazard ratios for the BioMonitor versus control group including 95% CI are additionally calculated based on the Cox regression model for the following conditions:

- ITT analysis set, uncorrected adjudication, stratification amikind\_multi= STEMI/NSTEMI
- ITT analysis set, corrected adjudication,
- stratification amikind\_multi= STEMI/NSTEMI
- ITT analysis set, corrected adjudication,
- without stratification
- PP analysis set, corrected adjudication,
- stratification amikind\_multi= STEMI/NSTEMI
- PP analysis set, corrected adjudication,
- without stratification

The assumption of proportional hazards is checked graphically by log-minus-log survival versus log-time plots.



# 12. Sec. Endpoint: Time to 1st arrhythmia detection

#### 12.1. Analysis set

This endpoint is analyzed exclusively for the final statistical analysis report based on the ITT analysis set.<sup>79</sup>

#### 12.2. Variables

#### <u>CIP Chapter 8.3.2 Secondary endpoint: Time to first arrhythmia detection</u>

This secondary endpoint comprises the time from randomization to the detection of an arrhythmia that requires guideline-recommended therapy. Patients without arrhythmia detection are censored, i.e. the time from randomization until the earliest date of drop-out, study termination, or date of freezing the Clinical Data Management System database (in case of interim analyses) is considered.

To be more precise, secondary endpoints will not be analyzed during interim analyzes and the earliest date of drop-out is just documented as termination date date\_term at the termination CRF.

| Data file:Identifier record id | Notes | Variable<br>name | L 1 1 1 1 1 | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| advers_events | No<br>report | arr_date | When was the earliest documentation of the arrhythmia? | date | n.a. |
| adverse_events | No<br>report | arr_yn | Was an arrhythmia documented in the context of this event? | nominal | Yes / No |
| adverse_events | No<br>report | arrchange_yn | Does the arrhythmia require guideline-<br>recommended change of therapy? | nominal | Yes / No |
| data_ae_SAR | No<br>report | arrdetect_SAR <sup>80</sup> | | nominal | Yes / No |
| data_ae_SAR | No<br>report | | Date of a arrhythmia detection with guideline-<br>recommended change of therapy | date | n.a. |



| Data file: Identifier patient_display_id_full | | | l | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| data_SAR | descr. | | Any arrhythmia with guideline-<br>recommended change of therapy after<br>effective randomization ITT | nominal | Yes / No |
| data_SAR | No<br>report | | Date of 1st arrhythmia with guideline-<br>recommended change of therapy after<br>effective randomization ITT | date | n.a. |
| data_SAR | descr. | _SAR <sup>84</sup> | Days from effective randomization to 1st arrhythmia detection with guideline recommended therapy or termination ITT | scale | n.a. |

Spurious data, which were not clarified by the query process before CDMS closure, are indicated. If appropriate, descriptive and inferential analyses are performed both with /without such data.

#### 12.4. Exclusion of Particular Information

No data from the previous defined analysis set are excluded from the analysis except those defined in chapter 5.5, if applicable.

#### 12.5. Descriptive Analyses

If applicable, mean and median survival times are presented by using the Kaplan-Meier estimates. Kaplan-Meier survival figures are presented for illustration.

Other descriptive data will be presented via tables as specified in chapter 5.1.

#### 12.6. Hypotheses & Statistical Tests

#### CIP Chapter 7.3 Secondary hypotheses

The objective to show that arrhythmias requiring guideline-recommended therapy will be detected earlier in the BioMonitor group will be formally tested similarly to the primary hypothesis. The HR is defined as the rate of the BioMonitor group divided by the rate of the control group.

 $H_0$ : Null hypothesis:  $H_0$ :  $HR \le 1$  which means that monitoring patients of the BioMonitor group will not lead to a shorter time to first arrhythmia that requires guideline-recommended therapy, in the BioMonitor group compared to the control group.

 $H_A$ : Alternative hypothesis:  $H_A$ : HR >1 which means that monitoring patients of the BioMonitor group will lead to a shorter time to first arrhythmia that requires guideline-recommended therapy compared to the control group.



### 13. Other sec. EP: Time to all-cause death or heart transpl.

#### 13.1. Analysis set

This endpoint is analyzed exclusively for the final statistical analysis report based on the ITT analysis set.<sup>85</sup>

#### 13.2. Variables

#### <u>CIP Chapter 8.3.3.1. Time to death from any cause or heart transplantation</u>

Assessment of the time from randomization to death for any reason or heart transplantation during the clinical investigation.

| Data file: Identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_ | | name | label | level | values |
| display_id_full | | | | | |
| data_SAR | descr. | death_htx_ITT_SAR <sup>86</sup> | Death or heart transplantation ITT | nominal | Yes / No |
| | | | · | | |
| data_SAR | descr. | days_effrand_to_term_ | Days from effective randomization to | scale | n.a. |
| | | ITT_SAR <sup>87</sup> | termination ITT | | |

#### 13.3. Treatment of Missing and Spurious Data

Spurious data, which were not clarified by the query process before CDMS closure, are indicated. If appropriate, descriptive and inferential analyses are performed both with /without such data.

#### 13.1. Exclusion of Particular Information

No data from the previous defined analysis set are excluded from the analysis except those defined in chapter 5.5, if applicable.

#### 13.2. Descriptive Analyses

If applicable, mean and median survival times are presented by using the Kaplan-Meier estimates. Kaplan-Meier survival figures are presented for illustration.

Other descriptive data will be presented via tables as specified in chapter 5.1.

#### 13.1. Hypotheses & Statistical Tests



### 14. Other sec. EP: Time to CV death or heart transplantation

#### 14.1. Analysis set

This endpoint is analyzed exclusively for the final statistical analysis report based on the ITT analysis set.<sup>88</sup>

#### 14.2. Variables

#### CIP Chapter 8.3.3.2 Time to cardiovascular death or heart transplantation

Assessment of the time from randomization to cardiovascular death or heart transplantation during the clinical investigation. A specified endpoint definition will be given by the members of the EAEC ...

| Data file: Identifier patient_display_id_full | | Variable<br>name | | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| data_SAR | descr. | cvdeath_htx_ITT_SAR <sup>89</sup> | CV death or heart transplantation ITT | nominal | Yes / No |
| data_SAR | descr. | | Days from effective randomization to termination ITT | scale | n.a. |

#### 14.3. Treatment of Missing and Spurious Data

Spurious data, which were not clarified by the query process before CDMS closure, are indicated. If appropriate, descriptive and inferential analyses are performed both with /without such data.

#### 14.4. Exclusion of Particular Information

No data from the previous defined analysis set are excluded from the analysis except those defined in chapter 5.5, if applicable.

#### 14.5. Descriptive Analyses

If applicable, mean and median survival times are presented by using the Kaplan-Meier estimates. Kaplan-Meier survival figures are presented for illustration.

Other descriptive data will be presented via tables as specified in chapter 5.1.

#### 14.6. Hypotheses & Statistical Tests

Differences of the survival curves BioMonitor versus control group are tested for statistical inference with the log-rank test.



# 15. Other sec. EP: Time to 1<sup>st</sup> worsening of the patient status due to heart failure ...

#### 15.1. Analysis set

This endpoint is analyzed exclusively for the final statistical analysis report based on the ITT analysis set. $^{91}$ 

#### 15.2. Variables

<u>CIP Chapter 8.3.3.3 Time to first worsening of the patient status due to heart failure requiring hospitalization or urgent visit</u>

Assessment of the time from randomization to first hospitalization or urgent visit for worsening of the patient status due to heart failure, or death due to heart failure. A specified endpoint definition will be given by the members of the EAEC and documented in the charter agreement

| Data file: Identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient | Notes | | l | | values |
| display id full | | | label | levei | values |
| data SAR | doscr | any hf ITT SAR <sup>92</sup> | Any hospitalization or urgent visit for | nominal | Yes / No |
| uata_SAIN | uesci. | , , = = = | worsening of the patient status due to | Hommai | 163 / 140 |
| | | 1 | , , | | |
| | | 1 | heart failure, or death due to heart | | |
| | | | failure after effective randomization ITT | | |
| data_SAR | No | date_1hf_ITT_SAR <sup>93</sup> | Date of 1st hospitalization or urgent visit | date | n.a. |
| | report | | for worsening of the patient status due to | | |
| | | | heart failure, or death due to heart | | |
| | | | failure after effective randomization ITT | | |
| data_SAR | descr. | days_effrand_to_1hf_ITT_SAR <sup>94</sup> | Days from effective randomization to 1st <sup>t</sup> | scale | n.a. |
| | | | hospitalization or urgent visit for | | |
| | | | worsening of the patient status due to | | |
| | | | heart failure, or death due to heart | | |
| | | | failure or termination ITT | | |



Spurious data, which were not clarified by the query process before CDMS closure, are indicated. If appropriate, descriptive and inferential analyses are performed both with /without such data.

#### 15.1. Exclusion of Particular Information

No data from the previous defined analysis set are excluded from the analysis except those defined in chapter 5.5, if applicable.

#### 15.2. Descriptive Analyses

If applicable, mean and median survival times are presented by using the Kaplan-Meier estimates. Kaplan-Meier survival figures are presented for illustration.

Other descriptive data will be presented via tables as specified in chapter 5.1.

#### 15.3. Hypotheses & Statistical Tests

Differences of the survival curves BioMonitor versus control group are tested for statistical inference with the log-rank test.



# 16. Other sec. EP: Time to 1<sup>st</sup> hosp. resulting from an arrhythmia

#### 16.1. Analysis set

This endpoint is analyzed exclusively for the final statistical analysis report based on the ITT analysis set.<sup>95</sup>

#### 16.2. Variables

CIP chapter 8.3.3.4. Time to first hospitalization resulting from an arrhythmia Assessment of the time from randomization to the first hospitalization resulting from an arrhythmia or death resulting from arrhythmia. A specified endpoint definition will be given by the members of the EAEC and documented in the charter agreement.

| Data file: Identifier patient_display_id_full | | name | | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| data_SAR | descr. | any_arr_ITT_SAR <sup>96</sup> | Any hospitalization resulting from an arrhythmia or death resulting from arrhythmia after effective randomization ITT | nominal | Yes / No |
| data_SAR | No<br>report | date_1arr_ITT_SAR <sup>97</sup> | Date of 1st hospitalization resulting from an arrhythmia or death resulting from arrhythmia after effective randomization ITT | date | n.a. |
| data_SAR | descr. | ' | Days from effective randomization to 1st hospitalization resulting from an arrhythmia or death resulting from arrhythmia or termination ITT | scale | n.a. |





Spurious data, which were not clarified by the query process before CDMS closure, are indicated. If appropriate, descriptive and inferential analyses are performed both with /without such data.

#### 16.1. Exclusion of Particular Information

No data from the previous defined analysis set are excluded from the analysis except those defined in chapter 5.5, if applicable.

#### 16.2. Descriptive Analyses

If applicable, mean and median survival times are presented by using the Kaplan-Meier estimates. Kaplan-Meier survival figures are presented for illustration.

Other descriptive data will be presented via tables as specified in chapter 5.1.

#### 16.3. Hypotheses & Statistical Tests

Differences of the survival curves BioMonitor versus control group are tested for statistical inference with the log-rank test.



# 17. Other sec. EP: Time to 1<sup>st</sup> hosp. resulting from acute coronary syndrome

#### 17.1. Analysis set

This endpoint is analyzed exclusively for the final statistical analysis report based on the ITT analysis set.  $^{99}$ 

#### 17.2. Variables

<u>CIP cChapter 8.3.3.5. Time to first hospitalization resulting from acute coronary syndrome</u>

Assessment of the time from randomization to the first hospitalization resulting from acute coronary syndrome or death resulting from acute coronary syndrome. A specified endpoint definition will be given by the members of the EAEC and documented in the charter agreement.

| Data file: Identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_ | | name | label | level | values |
| display_id_full | | | | | |
| data_SAR | descr. | any_acs_ITT_SAR <sup>100</sup> | Any hospitalization resulting from acute | nominal | Yes / No |
| | | | coronary syndrome or death resulting | | |
| | | | from acute coronary syndrome after | | |
| | | | effective randomization ITT | | |
| data_SAR | No | date_1acs_ITT_SAR <sup>101</sup> | Date of 1st hospitalization resulting | date | n.a. |
| | report | | from acute coronary syndrome or death | | |
| | | | resulting from acute coronary | | |
| | | | syndrome after effective randomization | | |
| | | | ITT | | |
| data_SAR | descr. | days_effrand_to_1acs_ITT_SAR <sup>102</sup> | Days from effective randomization to | scale | n.a. |
| | | | 1st hospitalization resulting from acute | | |
| | | | coronary syndrome or death resulting | | |
| | | | from acute coronary syndrome or | | |
| | | | termination ITT | | |





Spurious data, which were not clarified by the query process before CDMS closure, are indicated. If appropriate, descriptive and inferential analyses are performed both with /without such data.

#### 17.1. Exclusion of Particular Information

No data from the previous defined analysis set are excluded from the analysis except those defined in chapter 5.5, if applicable.

#### 17.2. Descriptive Analyses

If applicable, mean and median survival times are presented by using the Kaplan-Meier estimates. Kaplan-Meier survival figures are presented for illustration.

Other descriptive data will be presented via tables as specified in chapter 5.1.

#### 17.3. Hypotheses & Statistical Tests

Differences of the survival curves BioMonitor versus control group are tested for statistical inference with the log-rank test.



# 18. Other sec. EP: Time to 1st hosp. resulting from stroke

#### 18.1. Analysis set

This endpoint is analyzed exclusively for the final statistical analysis report based on the ITT analysis set.  $^{103}$ 

#### 18.2. Variables

#### CIP Chapter 8.3.3.6 Time to first hospitalization resulting from stroke

Assessment of the time from randomization to the first hospitalization resulting from stroke or death resulting from stroke. A specified endpoint definition will be given by the members of the EAEC and documented in the charter agreement.

| Data file: Identifier patient_display_id_full | | Variable<br>name | | | Nominal<br>values |
|---|---|---|---|---|---|
| data_SAR | descr. | any_stroke_ITT_SAR <sup>104</sup> | Any hospitalization resulting from stroke or death resulting from stroke after effective randomization ITT | nominal | Yes / No |
| data_SAR | No<br>report | date_1stroke_ITT_SAR <sup>105</sup> | Date of 1st hospitalization resulting from stroke or death resulting from stroke after effective randomization ITT | date | n.a. |
| data_SAR | descr. | 106 | Days from effective randomization to<br>the 1st hospitalization resulting from<br>stroke or death resulting from stroke<br>or termination ITT | scale | n.a. |





Spurious data, which were not clarified by the query process before CDMS closure, are indicated. If appropriate, descriptive and inferential analyses are performed both with /without such data.

#### 18.1. Exclusion of Particular Information

No data from the previous defined analysis set are excluded from the analysis except those defined in chapter 5.5, if applicable.

#### 18.2. Descriptive Analyses

If applicable, mean and median survival times are presented by using the Kaplan-Meier estimates. Kaplan-Meier survival figures are presented for illustration.

Other descriptive data will be presented via tables as specified in chapter 5.1.

#### 18.3. Hypotheses & Statistical Tests

Differences of the survival curves BioMonitor versus control group are tested for statistical inference with the log-rank test.



# 19. Other sec. EP: Time to 1<sup>st</sup> hosp. resulting from major bleeding

#### 19.1. Analysis set

This endpoint is analyzed exclusively for the final statistical analysis report based on the ITT analysis set.  $^{107}$ 

#### 19.2. Variables

CIP Chapter 8.3.3.7 Time to first hospitalization resulting from major bleeding

Assessment of the time from randomization to the first hospitalization resulting from major bleeding or death resulting from major bleeding. A specified endpoint definition will be given by the members of the EAEC and documented in the charter agreement.

| Data file: Identifier patient_display_id_full | | name | 1. 1. 1. 1. 1. | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| data_SAR | descr. | any_bleed_ITT_SAR <sup>108</sup> | Any hospitalization resulting from major bleeding or death resulting from major bleeding after effective randomization ITT | nominal | Yes / No |
| data_SAR | No<br>report | date_1bleed_ITT_SAR <sup>109</sup> | Date of 1st hospitalization resulting from<br>major bleeding or death resulting from<br>major bleeding after effective<br>randomization ITT | date | n.a. |
| data_SAR | | SAR <sup>110</sup> | Days from effective randomization to 1st hospitalization resulting from major bleeding or death resulting from major bleeding or termination ITT | scale | n.a. |





Spurious data, which were not clarified by the query process before CDMS closure, are indicated. If appropriate, descriptive and inferential analyses are performed both with /without such data.

#### 19.1. Exclusion of Particular Information

No data from the previous defined analysis set are excluded from the analysis except those defined in chapter 5.5, if applicable.

#### 19.2. Descriptive Analyses

If applicable, mean and median survival times are presented by using the Kaplan-Meier estimates. Kaplan-Meier survival figures are presented for illustration.

Other descriptive data will be presented via tables as specified in chapter 5.1.

#### 19.3. Hypotheses & Statistical Tests

Differences of the survival curves BioMonitor versus control group are tested for statistical inference with the log-rank test.



# 20. Other sec. EP: Time to 1<sup>st</sup> hosp. resulting from systemic embolism

#### 20.1. Analysis set

This endpoint is analyzed exclusively for the final statistical analysis report based on the ITT analysis set. $^{111}$ 

#### 20.2. Variables

CIP Chapter 8.3.3.8 Time to first hospitalization resulting from systemic embolism

Assessment of the time from randomization to the first hospitalization resulting from systemic embolism or death resulting from systemic embolism. A specified endpoint definition will be given by the members of the EAEC and documented in the charter agreement.

| Data file: Identifier patient_display_id_full | Notes | | | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| data_SAR | descr. | , | Any hospitalization resulting from systemic embolism or death resulting from systemic embolism. after effective randomization ITT | nominal | Yes / No |
| data_SAR | No<br>report | | Date of 1st hospitalization resulting from systemic embolism or death resulting from systemic embolism. after effective randomization ITT | date | n.a. |
| data_SAR | | SAR <sup>114</sup> | Days from effective randomization to 1st hospitalization resulting from systemic embolism or death resulting from systemic embolism or termination ITT | scale | n.a. |





Spurious data, which were not clarified by the query process before CDMS closure, are indicated. If appropriate, descriptive and inferential analyses are performed both with /without such data.

#### 20.1. Exclusion of Particular Information

No data from the previous defined analysis set are excluded from the analysis except those defined in chapter 5.5, if applicable.

#### 20.2. Descriptive Analyses

If applicable, mean and median survival times are presented by using the Kaplan-Meier estimates. Kaplan-Meier survival figures are presented for illustration.

Other descriptive data will be presented via tables as specified in chapter 5.1.

#### 20.3. Hypotheses & Statistical Tests

Differences of the survival curves BioMonitor versus control group are tested for statistical inference with the log-rank test.



# 21. Other sec. EP: Time to 1<sup>st</sup> arrhythmia

#### 21.1. Analysis set

This endpoint is analyzed exclusively for the final statistical analysis report based on the ITT analysis set. $^{115}$ 

#### 21.2. Variables

#### CIP Chapter 8.3.3.9. Time to first arrhythmia

Assessment of the time from randomization to first arrhythmia.

| Data file: Identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| record_ID | | name | label | level | values |
| adverse_events | No | arr_yn | NEW: Arrhythmia documented | nominal | Yes / No |
| | report | | | | |
| advers_events | No | arr_date | NEW: Earliest documentation | date | n.a. |
| | report | | of the arrhythmia | | |
| adverse_events | No | end_date | End date of AE | date | n.a. |
| | report | | (if applicable: Date of death) | | |

| Data file: Identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_display_id_full | | name | label | level | values |
| data_SAR | No | any_arrhythmia_ITT_SAR <sup>116</sup> | Any arrhythmia after effective | nominal | Yes / No |
| | report | | randomization ITT | | |
| data_SAR | No | date_1arrhythmia_ITT_SAR <sup>117</sup> | Date of 1st arrhythmia after | date | n.a. |
| | report | - | effective randomization ITT | | |
| data_SAR | descr. | days_effrand_to_1arrhythmia_ | Days from effective | scale | n.a. |
| | | ITT_SAR <sup>118</sup> | randomization to 1st | | |
| | | | arrhythmia or termination ITT | | |





Spurious data, which were not clarified by the query process before CDMS closure, are indicated. If appropriate, descriptive and inferential analyses are performed both with /without such data.

#### 21.1. Exclusion of Particular Information

No data from the previous defined analysis set are excluded from the analysis except those defined in chapter 5.5, if applicable.

#### 21.2. Descriptive Analyses

If applicable, mean and median survival times are presented by using the Kaplan-Meier estimates. Kaplan-Meier survival figures are presented for illustration.

Other descriptive data will be presented via tables as specified in chapter 5.1.

#### 21.3. Hypotheses & Statistical Tests

Differences of the survival curves BioMonitor versus control group are tested for statistical inference with the log-rank test.



### 22. Other sec. EP: Type of initiated therapies

The main objective of this endpoint is to describe in an exploratorive fashion which therapies are introduced to patients as consequence of BioMonitor detected arrhythmias. Therefore an internal adjudication board classified the information given in text entries of relevant AE reports with respect to cardiac rhythm, initiated or changed drug therapy, and initiated device therapy.

#### 22.1. Analysis set

This endpoint is analyzed exclusively for the final statistical analysis report based on the ITT analysis set. 119

#### 22.2. Variables

CIP Chapter 8.3.3.10 Type of initiated therapies.

Evaluation of the diagnoses and consequent type of therapies based on ICM-detected arrhythmias.

| | | | | | · | |
|---|---|---|---|---|---|---|
| Data file: Identifier parent_record_id (related to the AE record ID) | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal | values |
| internal_adjudication | *# | adj_rhythm_multi | · | | Atrial fibrillation Atrial flutter AV block Bradycardia frequent VPBs non-sustained VT sustained VT polymorphic VT/VF Other SVT Pause None | |
| internal_adjudication | descriptive<br>* | adj_drug | Drug | | Antiarrhythmic<br>BB<br>Diuretic<br>OAC<br>Other<br>None | |
| internal_adjudication | Case listing | adj_drug_txt | Drug text | text | n.a. | |
| internal_adjudication | | adj_device | Device | nominal | Ablation<br>Cardioversion<br>ICD<br>Other<br>PM<br>None | |
| internal_adjudication | Case listing | adj_device_txt | Device text | text | n.a. | |

<sup>\*2</sup>x3 contingency table; # 2x3 contingency table



<sup>&</sup>lt;sup>119</sup> analysis\_set\_itt\_SAR = Yes

Spurious data, which were not clarified by the query process before CDMS closure, are indicated. If appropriate, descriptive and inferential analyses are performed both with /without such data.

#### 22.1. Exclusion of Particular Information

No data from the previous defined analysis set are excluded from the analysis except those defined in chapter 5.5, if applicable.

#### 22.2. Descriptive Analyses

Descriptive data are presented via tables as specified in chapter 5.1.

#### 22.3. Hypotheses & Statistical Tests

A broad range of diagnoses and therapies can be expected for the study population. A reasonable pre-defined scheme to classify the events has not yet been developed. Thus, there are no pre-specified statistical tests for this endpoint.



## 23. Other sec. EP: Time to 1st therapy.

#### 23.1. Analysis set

This endpoint is analyzed exclusively for the final statistical analysis report based on the ITT analysis set. $^{120}$ 

#### 23.2. Variables

#### CIP Chapter 8.3.3.11 Time to 1st therapy

Assessment of the time from randomization to first therapy. In this context therapy is the attempted remediation of the patient's regular heartbeat. To ensure a standardized proceeding, guideline-based therapy recommendations will be provided to the participating investigators within a separate manual.

This endpoint comprises therapies reported in AE report CRF, irrespective of the cause of the patient being in the investigational site. The patient may be called in by an investigator after arrhythmias were detected in the BM or after a physician outside the investigational site assumed it appropriate to send the patient to a highly competent cardiological site. Changes of therapy prescribed by a general practitioner or another physician outside the investigational site are not considered.

Since the investigational sites are highly specialized cardiological units, it is not assumed that they will prescribe a relevant amount of non-cardiovascular therapies. All cardiovascular therapies will be considered for this endpoint, also if they are not directly relevant for the regular heartbeat as stated in the CIP. Especially, this also includes therapies directed at diuresis, blood pressure, coagulation status or ischemia, since all these treatments do also interact with the heart rhythm in some way.

| Data file: Identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| record_id | | name | label | level | values |
| general_notification | No<br>report | visit_date | Date of patient visit in investigational site | date | n.a. |
| general_notification_<br>data_SAR | No<br>report | 1 7 = 3 = | Date of the guideline-recommended change of therapy after an AE | date | n.a. |

| Data file: Identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| record_id | | name | label | level | values |
| arrhythmia_notification | No | visit_date | Date of patient visit in investigational site | date | n.a. |
| | report | | | | |
| arrhythmia_notification_ | No | therapy_arr_date | Date of the guideline-recommended change | date | n.a. |
| data_SAR | report | . , _ | of therapy after an AE | | |

| Data file: Identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| record_id | | name | label | level | values |
| · · · · · - · | No<br>report | | NEW: Record ID of the parent document, i.e.<br>the general notification CRF or arrhythmia<br>notification CRF related to the AE CRF | nominal | |
| adverse_events | No<br>report | | Does the arrhythmia require guideline-<br>recommended change of therapy | nominal | Yes / No |



<sup>&</sup>lt;sup>120</sup> analysis\_set\_itt\_SAR = Yes

| Data file: Identifier patient_display_id_full | Notes | Variable name | | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| data_SAR | No<br>report | any_therapy_ITT_SAR <sup>121</sup> | Any therapy after effective randomization (attempted remediation of the patient's regular heartbeat) ITT | nominal | Yes / No |
| data_SAR | No<br>report | date_1therapy_ITT_SAR | Date of 1st therapy (attempted remediation of the patient's regular heartbeat) ITT | date | n.a. |
| data_SAR | descr. | 1therapy_ITT_SAR <sup>123</sup> | Days from randomization to 1st therapy (attempted remediation of the patient's regular heartbeat) or termination ITT | scale | n.a. |

Spurious data, which were not clarified by the query process before CDMS closure, are indicated. If appropriate, descriptive and inferential analyses are performed both with /without such data.

#### 23.1. Exclusion of Particular Information

No data from the previous defined analysis set are excluded from the analysis except those defined in chapter 5.5, if applicable.

#### 23.2. Descriptive Analyses

If applicable, mean and median survival times are presented by using the Kaplan-Meier estimates. Kaplan-Meier survival figures are presented for illustration.

Other descriptive data will be presented via tables as specified in chapter 5.1.

#### 23.3. Hypotheses & Statistical Tests

Differences of the survival curves BioMonitor versus control group are tested for statistical inference with the log-rank test.



### 24. Other sec. EP: Quality of Life / WHO-5 Well-being Index

#### 24.1. Analysis set

This endpoint is analyzed exclusively for the final statistical analysis report based on the ITT analysis set. 124

#### 24.2. Variables

#### CIP Chapter 8.3.3.12 Quality of Life (QoL)

A further secondary endpoint is the assessment of the patient's quality of life. The patient's quality of life will be recorded during the regular telephone contacts using the WHO-5 Wellbeing Index.

| Data file: Identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| record_ID | | name | label | level | values |
| who_five_<br>well_being_index | | interview_<br>interval | Interval (filled in automatically) | | 1. Quality of Life (6 M) 2. Quality of Life (12 M) 3. Quality of Life (18 M) 4. Quality of Life (24 M) 5. Quality of Life (30 M) 6. Quality of Life (36 M) 7. Quality of Life (42 M) 8. Quality of Life (48 M) 9. Quality of Life (54 M) 10. Quality of Life (60 M) |
| | | q1_multi | I have felt cheerful and good spirits | ordinal | 0,1,2,3,4,5 |
| | i | q2_multi | I have felt calm and relaxed | ordinal | 0,1,2,3,4,5 |
| | | q3_multi | I have felt active and vigorous | ordinal | 0,1,2,3,4,5 |
| | | q4_multi | | ordinal | 0,1,2,3,4,5 |
| | | | My daily life has been filled with things<br>that interest me | ordinal | 0,1,2,3,4,5 |

| Data file: Identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_display_id_full | | name | label | level | values |
| data_SAR | descr. | wbi_percscore_6m_SAR <sup>125</sup> | WBI percentage score: 6m | scale | 0-100 |
| data_SAR | descr. | wbi_percscore_12m_SAR <sup>126</sup> | WBI percentage score: 12m | scale | 0-100 |
| data_SAR | descr. | wbi_percscore_18m_SAR <sup>127</sup> | WBI percentage score: 18m | scale | 0-100 |
| data_SAR | descr. | wbi_percscore_24m_SAR <sup>128</sup> | WBI percentage score: 24m | scale | 0-100 |
| data_SAR | descr. | wbi_percscore_30m_SAR <sup>129</sup> | WBI percentage score: 30m | scale | 0-100 |
| data_SAR | descr. | wbi_percscore_36m_SAR <sup>130</sup> | WBI percentage score: 36m | scale | 0-100 |
| data_SAR | descr. | wbi_percscore_42m_SAR <sup>131</sup> | WBI percentage score: 42m | scale | 0-100 |
| data_SAR | descr. | wbi_percscore_48m_SAR <sup>132</sup> | WBI percentage score: 48m | scale | 0-100 |
| data_SAR | descr. | wbi_percscore_54m_SAR <sup>133</sup> | WBI percentage score: 54m | scale | 0-100 |
| data_SAR | descr. | wbi_percscore_60m_SAR <sup>134</sup> | WBI percentage score: 60m | scale | 0-100 |
| data_SAR | descr. | wbi_percscore_24m_6m_SAR <sup>135</sup> | WBI percentage score: | scale | -100 till 100 |
| | | | Difference 24m vs. 6m | | |
| data_SAR | descr. | wbi_percscore_48m_6m_SAR <sup>136</sup> | WBI percentage score: | scale | -100 till 100 |
| | | | Difference 48m vs. 6m | | |

Spurious data, which were not clarified by the query process before CDMS closure, are indicated. If appropriate, descriptive and inferential analyses are performed both with /without such data.

Missing data from a specific in hospital follow-up is imputed with the Last-Observation-Carry-Forward method, i.e. data from the nearest previous in-hospital follow-up, if available.

#### 24.1. Exclusion of Particular Information

No data from the previous defined analysis set are excluded from the analysis except those defined in chapter 5.5, if applicable.

#### 24.2. Descriptive Analyses

Descriptive data are presented via tables as specified in chapter 5.1.

#### 24.3. Hypotheses & Statistical Tests

The percentage Well-Being Index for the 6m in-hospital FU, 24m in-hospital FU, 48m in-hospital FU, differences between 24m and 6m, and differences between 48m and 6m are analyzed BioMonitor versus control group with the Mann-Whitney-U test.





### 25. Data of Interest: Quality of Life / EQ-5D

#### 25.1. Analysis set

This endpoint is analyzed exclusively for the final statistical analysis report based on the ITT analysis set.  $^{137}$ 

#### 25.2. Variables

#### CIP Chapter 8.4 Further data of interest

In addition, the EQ-5D-5L questionnaire will be administered during the telephone contacts to estimate utility values at different time points for an economic evaluation.

| Data file:<br>Identifier<br>record_id | Notes | Variable<br>name | Variable<br>label | level | Nominal values |
|---|---|---|---|---|---|
| eq_5d_5l_<br>questionnaire | no<br>report | interval | in<br>automatically) | | 0. Quality of Life (Base) 1. Quality of Life (6 M) 2. Quality of Life (12 M) 3. Quality of Life (18 M) 4. Quality of Life (24 M) 5. Quality of Life (30 M) 6. Quality of Life (36 M) 7. Quality of Life (42 M) 8. Quality of Life (48 M) 9. Quality of Life (54 M) 10. Quality of Life (60 M) |
| | descr. | EQ5D5L_q1_mobility | MOBILITY | | slight problems walking<br>moderate problems walking<br>severe problems walking<br>unable to walk |
| | descr. | EQ5D5L_q2_selfcare | - SELF-CARE | | no problems washing or dressing yourself slight problems washing or dressing yourself moderate problems washing or dressing yourself severe problems washing or dressing yourself unable to wash or dress yourself |
| | descr. | activities | health TODAY – USUAL ACTIVITIES | nominal | no problems doing your usual activities slight problems doing your usual activities moderate problems doing your usual activities severe problems doing your usual activities unable to do your usual activities |
| | descr. | discomfort | - PAIN/<br>DISCOMFORT | | no pain or discomfort<br>slight pain or discomfort<br>moderate pain or discomfort<br>severe pain or discomfort<br>extreme pain or discomfort |
| | descr. | EQ5D5L_q5_anxiety<br>_depression | -ANXIETY /<br>DEPRESSION | nominal | not anxious or depressed<br>slightly anxious or depressed<br>moderately anxious or depressed<br>severely anxious or depressed<br>extremely anxious or depressed |
| | descr. | | Scale number indicating the respondent's health today' | metric | 0-100 |



| Data file: Identifier patient_display_id_full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| data_SAR | descr. | EQ5D5L_health_scale_bas_SAR <sup>138</sup> | EQ5D5L score: Baseline | scale | 0-100 |
| data_SAR | descr. | EQ5D5L_health_scale_6m_SAR <sup>139</sup> | EQ5D5L score: 6m | scale | 0-100 |
| data_SAR | descr. | EQ5D5L_health_scale_12m_SAR <sup>140</sup> | EQ5D5L score: 12m | scale | 0-100 |
| data_SAR | descr. | EQ5D5L_health_scale_18m_SAR <sup>141</sup> | EQ5D5L score: 18m | scale | 0-100 |
| data_SAR | descr. | EQ5D5L_health_scale_24m_SAR <sup>142</sup> | EQ5D5L score: 24m | scale | 0-100 |
| data_SAR | descr. | EQ5D5L_health_scale_30m_SAR <sup>143</sup> | EQ5D5L score: 30m | scale | 0-100 |
| data_SAR | descr. | EQ5D5L_health_scale_36m_SAR <sup>144</sup> | EQ5D5L score: 36m | scale | 0-100 |
| data_SAR | descr. | EQ5D5L_health_scale_42m_SAR <sup>145</sup> | EQ5D5L score: 42m | scale | 0-100 |
| data_SAR | descr. | EQ5D5L_health_scale_48m_SAR <sup>146</sup> | EQ5D5L score: 48m | scale | 0-100 |
| data_SAR | descr. | EQ5D5L_health_scale_54m_SAR <sup>147</sup> | EQ5D5L score: 54m | scale | 0-100 |
| data_SAR | descr. | EQ5D5L_health_scale60m_SAR <sup>148</sup> | EQ5D5L score: 60m | scale | 0-100 |

Spurious data, which were not clarified by the query process before CDMS closure, are indicated. If appropriate, descriptive and inferential analyses are performed both with /without such data.

#### 25.1. Exclusion of Particular Information

No data from the previous defined analysis set are excluded from the analysis except those defined in chapter 5.5, if applicable.

#### 25.2. Descriptive Analyses

Descriptive data are presented via tables as specified in chapter 5.1.

#### 25.3. Hypotheses & Statistical Tests

There are no pre-specified hypotheses.





#### **Abbreviations**

ADE Adverse Device Effect

AE Adverse Event AF Atrial Fibrillation

CDMS Clinical Data Management System

CI Confidence Interval
CIP Clinical Investigation Plan
CIR Clinical Investigation Report

CRF Case Report Form CV Cardio vascular

DSMB Data Safety Monitoring Board EAEC Endpoint and Adverse Event Board

ECG Electrocardiogram

FU Follow-up

SADE Serious Adverse Device Event

SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Statistical Analysis Report SOP Standard Operating Procedure

SD Standard Deviation

